CLINICAL TRIAL: NCT03823287
Title: A Phase III, Multicenter, Randomized, Double-Masked, Active Comparator-Controlled Study to Evaluate the Efficacy and Safety of Faricimab in Patients With Neovascular Age-Related Macular Degeneration (TENAYA)
Brief Title: A Study to Evaluate the Efficacy and Safety of Faricimab in Participants With Neovascular Age-Related Macular Degeneration (TENAYA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GR40306; 2018-002152-32 (EudraCT Number)
Record Dates: First submitted 2019-01-29; First posted 2019-01-30 (Actual); Results first posted 2022-05-04 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Wet Macular Degeneration
Keywords: AMD; nAMD; neovascular age-related macular degeneration; choroidal neovascularization secondary to age-related macular degeneration
MeSH Terms: conditions — Wet Macular Degeneration | interventions — faricimab; aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Faricimab (Experimental)
  Interventions: Drug: Faricimab; Procedure: Sham Procedure
- Aflibercept (Active Comparator)
  Interventions: Drug: Aflibercept; Procedure: Sham Procedure

INTERVENTIONS:
Drug: Faricimab — Faricimab will be administered by intravitreal injection into the study eye at intervals as specified in the study protocol.
  Other Names: VABYSMO™; RO6867461; RG7716
  Arms: Faricimab
Drug: Aflibercept — Aflibercept will be administered by intravitreal injection into the study eye once every 4 weeks for 3 consecutive months, followed by once every 8 weeks (Q8W).
  Other Names: Eylea
  Arms: Aflibercept
Procedure: Sham Procedure — The sham is a procedure that mimics an intravitreal injection, but involves the blunt end of an empty syringe (without a needle) being pressed against the anesthetized eye. It will be administered to participants in both treatments arms at applicable visits to maintain masking.

SUMMARY:
This study will evaluate the efficacy, safety, durability, and pharmacokinetics of faricimab administered at intervals as specified in the protocol, compared with aflibercept once every 8 weeks (Q8W), in participants with neovascular age-related macular degeneration (nAMD).

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naïve choroidal neovascularization (CNV) secondary to age-related macular degeneration (nAMD) in the study eye
* Ability to comply with the study protocol, in the investigator's judgment
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use acceptable contraceptive measures that result in failure rate <1% per year during the treatment period and for at least 3 months after the final dose of study treatment
* Other protocol-specified inclusion criteria may apply

Exclusion Criteria:

* Uncontrolled blood pressure, defined as systolic blood pressure >180 millimeters of mercury (mmHg) and/or diastolic blood pressure >100 mmHg while a patient is at rest on Day 1
* Pregnancy or breastfeeding, or intention to become pregnant during the study
* CNV due to causes other than AMD in the study eye
* Any history of macular pathology unrelated to AMD affecting vision or contributing to the presence of intraretinal or subretinal fluid in the study eye
* Any concurrent intraocular condition in the study eye that, in the opinion of the investigator, could either reduce the potential for visual improvement or require medical or surgical intervention during the study
* Uncontrolled glaucoma in the study eye
* Any prior or concomitant treatment for CNV or vitreomacular-interface abnormalities in the study eye
* Prior IVT administration of faricimab in either eye
* History of idiopathic or autoimmune-associated uveitis in either eye
* Active ocular inflammation or suspected or active ocular or periocular infection in either eye
* Other protocol-specified exclusion criteria may apply

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 671 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2020-10-26 (Actual); Study Completion 2022-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (161):
- United States (52):
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Barnet Dulaney Perkins Eye Center, Phoenix, Arizona
  - Retina Associates Southwest PC, Tucson, Arizona
  - Retinal Diagnostic Center, Campbell, California
  - The Retina Partners, Encino, California
  - Jacobs Retina center at the Shiley eye Institute UCSD, La Jolla, California
  - South Coast Retina Center, Long Beach, California
  - Southern CA Desert Retina Cons, Palm Desert, California
  - California Eye Specialists Medical group Inc., Pasadena, California
  - Retina Consultants, San Diego, Poway, California
  - Retina Consultants of Southern California, Redlands, California
  - University of California, Davis, Eye Center, Sacramento, California
  - Retina Consultants of Southern, Colorado Springs, Colorado
  - Retina Group of New England, New London, Connecticut
  - Rand Eye, Deerfield Beach, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - Retina Vitreous Assoc of FL, St. Petersburg, Florida
  - Northwestern Medical Group/Northwestern University, Chicago, Illinois
  - Retina Associates, Lenexa, Kansas
  - Johns Hopkins Med, Baltimore, Maryland
  - Retina Group of Washington, Chevy Chase, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Associated Retinal Consultants, Grand Rapids, Michigan
  - Midwest Vision Research Foundation, Chesterfield, Missouri
  - Retina Associates of St. Louis, Florissant, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - NJ Retina, Edison, New Jersey
  - Retina Associates of NJ, Teaneck, New Jersey
  - Long Is. Vitreoretinal Consult, Great Neck, New York
  - Ophthalmic Cons of Long Island, Oceanside, New York
  - Retina Assoc of Western NY, Rochester, New York
  - The Retina Consultants, Slingerlands, New York
  - Retina Vit Surgeons/Central NY, Syracuse, New York
  - Western Carolina Retinal Associate PA, Asheville, North Carolina
  - Char Eye Ear &Throat Assoc, Charlotte, North Carolina
  - Graystone Eye, Hickory, North Carolina
  - Carolina Eye Associates, Southern Pines, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Retina Northwest, Portland, Oregon
  - Mid Atlantic Retina - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Charleston Neuroscience Inst, Ladson, South Carolina
  - Black Hills Eye Institute, Rapid City, South Dakota
  - Charles Retina Institute, Germantown, Tennessee
  - Tennessee Retina PC., Nashville, Tennessee
  - Texas Retina Associates, Dallas, Texas
  - Retina & Vitreous of Texas, Houston, Texas
  - Retina Consultants of Texas, Houston, Texas
  - Valley Retina Institute P.A., McAllen, Texas
  - Rocky Mountain Retina, Salt Lake City, Utah
  - Spokane Eye Clinical Research, Spokane, Washington
- Canada (9):
  - Calgary Retina Consultants, Calgary, Alberta
  - University of British Columbia - Vancouver Coastal Health Authority, Vancouver, British Columbia
  - Ivey Eye Institute, London, Ontario
  - University of Ottawa Eye Institute, Ottawa, Ontario
  - Retina Institute of Ottawa, Ottawa, Ontario
  - Toronto Retina Institute, Toronto, Ontario
  - Unity Health Toronto, Toronto, Ontario
  - Institut De L'Oeil Des Laurentides, Boisbriand, Quebec
  - Michel Giunta Clinique Medical, Sherbrooke, Quebec
- Germany (3):
  - Universitätsklinikum Freiburg, Klinik für Augenheilkunde, Freiburg im Breisgau
  - Universitätsklinik Heidelberg, Heidelberg
  - Universitätsklinikum Tübingen, Tübingen
- Hungary (4):
  - Budapest Retina Associates Kft., Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Ganglion Medial Center, Pécs
  - Zala Megyei Kórház, Zalaegerszeg
- Israel (5):
  - Rambam Medical Center, Haifa
  - Hadassah MC, Jerusalem
  - Rabin MC, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky MC, Tel Aviv
- Italy (4):
  - Ospedale Clinicizzato SS Annunziata, Chieti, Abruzzo
  - Fondazione G.B. Bietti Per Lo Studio E La Ricerca in Oftalmologia-Presidio Ospedaliero Britannico, Rome, Lazio
  - Fondazione Irccs Ca' Granda Ospedale Maggiore Policlinico-Clinica Regina Elena, Milan, Lombardy
  - Azienda Ospedaliera di Perugia Ospedale S. Maria Della Misericordia, Perugia, Umbria
- Japan (41):
  - Chukyo Hospital, Aichi
  - Nagoya University Hospital, Aichi
  - Nagoya City University Hospital, Aichi
  - Aichi Medical University Hospital, Aichi
  - Daiyukai Daiichi Hospital, Aichi
  - Chiba University Hospital, Chiba
  - Toho University Sakura Medical Center, Chiba
  - Hayashi Eye Hospital, Fukuoka
  - Kurume University Hospital, Fukuoka
  - Southern TOHOKU Eye Clinic, Fukushima
  - Sapporo City General Hospital, Hokkaido
  - Hokkaido University Hospital, Hokkaido
  - Asahikawa Medical University Hospital, Hokkaido
  - Hyogo Prefectural Amagasaki General Medical Center (Hyogo AGMC), Hyōgo
  - Hyogo Medical University Hospital, Hyōgo
  - Kozawa eye hospital and diabetes center, Ibaraki
  - Kagawa University Hospital, Kagawa
  - Kagoshima University Hospital, Kagoshima
  - Ideta Eye Hospital, Kumamoto
  - Kyoto University Hospital, Kyoto
  - Mie University Hospital, Mie
  - Fukushima Medical University Hospital, Miyagi
  - University of Miyazaki Hospital, Miyazaki
  - Shinshu University Hospital, Nagano
  - Iida Municipal Hospital, Nagano
  - Japanese Red Cross Nagasaki Genbaku Hospital, Nagasaki
  - Nara Medical University Hospital, Nara
  - University of the Ryukyus Hospital, Okinawa
  - Kitano Hospital, Osaka
  - Osaka Metropolitan University Hospital, Osaka
  - Kansai Medical University Medical Center, Osaka
  - Kansai Medical University Hospital, Osaka
  - National Defense Medical College Hospital, Saitama
  - Shiga University Of Medical Science Hospital, Shiga
  - Tokushima University Hospital, Tokushima
  - Nihon University Hospital, Tokyo
  - Takeuchi eye clinic, Tokyo
  - Tokyo Women's Medical University Hospital, Tokyo
  - Kyorin University Hospital, Tokyo
  - Tokyo Medical University Hachioji Medical Center, Tokyo
  - Yamaguchi University Hospital, Yamaguchi
- Mexico (3):
  - Centro Oftalmológico Mira, S.C, Cuauhtémoc, Mexico CITY (federal District)
  - Macula Retina Consultores, México, Mexico CITY (federal District)
  - Montemayor & Asociados (Oftalmologos), Monterrey, Nuevo León
- Netherlands (2):
  - Het Oogziekenhuis Rotterdam, Rotterdam
  - ETZ Elisabeth, Tilburg
- Poland (7):
  - Szpital sw. Lukasza, Bielsko-Biala
  - Specjalistyczny O?rodek Okulistyczny Oculomedica, Bydgoszcz
  - Szpital Specjalistyczny nr 1, Bytom
  - Dobry Wzrok Sp Z O O, Gdansk
  - Gabinet Okulistyczny Prof Edward Wylegala, Katowice
  - Centrum Medyczne Dietla 19 Sp. Z O.O., Krakow
  - SPEKTRUM Osrodek Okulistyki Klinicznej, Wroclaw
- Russia (3):
  - FSBI ?Scientific Research Institute of Eye Diseases? of Russian Academy of medical Sciences, Moscow, Moscow Oblast
  - Medical Military Academy n.a S.M.Kirov, Saint Petersburg, Sankt-Peterburg
  - Clinics of Eye Diseases, LLC, Kazan', Tatarstan Republic
- Spain (8):
  - Hospital General de Catalunya, Sant Cugat del Vallès, Barcelona
  - Instituto Oftalmologico Gomez Ulla, Santiago de Compostela, LA Coruna
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Oftalvist Valencia, Burjassot, Valencia
  - Hospital dos de maig, Barcelona
  - Clinica Universitaria de Navarra, Madrid
  - Clinica Baviera, Madrid
- Switzerland (2):
  - Vista Klinik Ophthalmologische Klinik, Binningen
  - Stadtspital Triemli Ophthalmologische Klinik, Zurich
- Turkey (Türkiye) (3):
  - Ankara Baskent University Medical Faculty; Department of Ophthalmology, Ankara
  - Kocaeli Üniversitesi Tıp Fakültesi; Department of Ophthalmology, Kocaeli
  - Selcuk University Faculty of Medicine; Department Of Ophthalmology, Konya
- United Kingdom (15):
  - Bradford Royal Infirmary, Bradford
  - Bristol Eye Hospital, Bristol
  - University Hospital of Wales, Cardiff
  - Frimley Park Hospital, Frimley
  - Gloucestershire Royal Hospital, Gloucester
  - Hull Royal Infirmary, Hull
  - St James University Hospital, Leeds
  - Royal Liverpool University Hospital, Liverpool
  - Moorfields Eye Hospital NHS Foundation Trust, London
  - Royal Free Hospital, London
  - Manchester Royal Infirmary, Manchester
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Southampton General Hospital, Southampton
  - New Cross Hospital, Wolverhampton
  - The York Hospital, York

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Result] Khanani AM, Kotecha A, Chang A, Chen SJ, Chen Y, Guymer R, Heier JS, Holz FG, Iida T, Ives JA, Lim JI, Lin H, Michels S, Quezada Ruiz C, Schmidt-Erfurth U, Silverman D, Singh R, Swaminathan B, Willis JR, Tadayoni R; TENAYA and LUCERNE Investigators. TENAYA and LUCERNE: Two-Year Results from the Phase 3 Neovascular Age-Related Macular Degeneration Trials of Faricimab with Treat-and-Extend Dosing in Year 2. Ophthalmology. 2024 Aug;131(8):914-926. doi: 10.1016/j.ophtha.2024.02.014. Epub 2024 Feb 19. PMID 38382813
- [Derived] Takahashi K, Cheung CMG, Iida T, Lai TYY, Ohji M, Yanagi Y, Kawano M, Ohsawa S, Suzuki T, Kotecha A, Lin H, Patel V, Swaminathan B, Lee WK; TENAYA, LUCERNE Investigators. Efficacy, durability, and safety of faricimab in patients from Asian countries with neovascular age-related macular degeneration: 1-Year subgroup analysis of the TENAYA and LUCERNE trials. Graefes Arch Clin Exp Ophthalmol. 2023 Nov;261(11):3125-3137. doi: 10.1007/s00417-023-06071-8. Epub 2023 Jun 9. PMID 37294433
- [Derived] Khanani AM, Guymer RH, Basu K, Boston H, Heier JS, Korobelnik JF, Kotecha A, Lin H, Silverman D, Swaminathan B, Willis JR, Yoon YH, Quezada-Ruiz C. TENAYA and LUCERNE: Rationale and Design for the Phase 3 Clinical Trials of Faricimab for Neovascular Age-Related Macular Degeneration. Ophthalmol Sci. 2021 Nov 17;1(4):100076. doi: 10.1016/j.xops.2021.100076. eCollection 2021 Dec. PMID 36246941
- [Derived] Heier JS, Khanani AM, Quezada Ruiz C, Basu K, Ferrone PJ, Brittain C, Figueroa MS, Lin H, Holz FG, Patel V, Lai TYY, Silverman D, Regillo C, Swaminathan B, Viola F, Cheung CMG, Wong TY; TENAYA and LUCERNE Investigators. Efficacy, durability, and safety of intravitreal faricimab up to every 16 weeks for neovascular age-related macular degeneration (TENAYA and LUCERNE): two randomised, double-masked, phase 3, non-inferiority trials. Lancet. 2022 Feb 19;399(10326):729-740. doi: 10.1016/S0140-6736(22)00010-1. Epub 2022 Jan 24. PMID 35085502

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 989 patients were screened, 318 of whom failed screening most commonly due to not meeting inclusion criteria. A total of 671 treatment-naive patients with nAMD were randomized 1:1 into the study: 334 to the faricimab arm and 337 to the aflibercept arm.
Groups:
- Arm A: Faricimab: Participants randomized to Arm A received 6 mg of faricimab intravitreally (IVT) once every 4 weeks (Q4W) up to Week 12 (4 injections). At Week 20, protocol-defined assessment of disease activity required Arm A participants with active disease to be treated with a once every 8 weeks (Q8W) dosing regimen of 6 mg of faricimab (i.e., injections at Weeks 20, 28, 36, 44, 52, and 60). A second protocol-defined assessment of disease activity at Week 24 required Arm A participants with active disease (excluding those with active disease at Week 20) to be treated with a once every 12 weeks (Q12W) dosing regimen of 6 mg of faricimab IVT (i.e., injections at Weeks 24, 36, 48, and 60). Participants receiving faricimab who did not have active disease according to the protocol-defined criteria at Week 20 and Week 24 were treated with 6 mg of faricimab IVT once every 16 weeks (Q16W) (i.e., injections at Weeks 28, 44, and 60). From Week 60 (when all Arm A participants were scheduled to receive study drug) to Week 108, Arm A participants were to be treated according to a personalized treatment interval (PTI) dosing regimen (Q8W, Q12W, or Q16W).
- Arm B: Aflibercept: Participants randomized to the active comparator (Arm B), a 2 mg dose of aflibercept was administered intravitreally (IVT) Q8W after 3 consecutive monthly doses during the 108-week treatment period. Participants were to receive 15 IVT injections of aflibercept during the 108-week treatment period. This will consist of three initiating injections (2 mg of aflibercept Q4W to Week 8), followed by 12 maintenance injections (2 mg of aflibercept Q8W at Weeks 16, 24, 32, 40, 48, 56, 64, 72, 80, 88, 96, and 104).
Period: Overall Study
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Started (Intent-to-Treat (ITT) Population) | 334 | 337
Received at Least One Dose of Study Drug (Safety Population) | 333 | 336
Completed up to Week 48 (Primary Completion Date Cutoff) | 319 | 323
Completed | 274 | 291
Not Completed | 60 | 46
Not completed — Withdrawal by Subject | 25 | 17
Not completed — Death | 13 | 7
Not completed — Lost to Follow-up | 7 | 8
Not completed — Adverse Event | 6 | 8
Not completed — Physician Decision | 5 | 2
Not completed — Lack of Efficacy | 2 | 0
Not completed — Other | 2 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept | Total
Number analyzed (Participants) | 334 | 337 | 671
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.9 (8.6) | 76.7 (8.8) | 76.3 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 191 | 211 | 402
  Male | 143 | 126 | 269
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 26 | 52
  Not Hispanic or Latino | 303 | 308 | 611
  Unknown or Not Reported | 5 | 3 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 303 | 302 | 605
  Asian | 26 | 28 | 54
  Black or African American | 0 | 3 | 3
  American Indian or Alaska Native | 1 | 2 | 3
  Multiple | 1 | 0 | 1
  Unknown | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States and Canada | 182 | 184 | 366
  Asia | 26 | 26 | 52
  Rest of the World | 126 | 127 | 253
Number of Participants by the Eye (Right or Left) Chosen as the Study Eye [Count of Participants; unit: Participants]
  Right Eye | 166 | 178 | 344
  Left Eye | 168 | 159 | 327
Best Corrected Visual Acuity (BCVA) Letter Score in the Study Eye [Mean (Standard Deviation); unit: ETDRS Letters] — Best corrected visual acuity (BCVA) at a starting test distance of 4 meters was measured using a set of three Precision VisionTM or Lighthouse distance acuity charts (modified ETDRS Charts 1, 2, and R). The BCVA letter score ranges from 0 to 100 (best score attainable), with a higher score indicating better visual acuity.
  ETDRS Letters | 61.3 (12.5) | 61.5 (12.9) | 61.4 (12.7)
Number of Participants by the BCVA Letter Score Categories in the Study Eye [Count of Participants; unit: Participants]
  ≥74 Letters | 47 | 52 | 99
  73 to 55 Letters | 200 | 201 | 401
  ≤54 Letters | 87 | 84 | 171
Number of Participants by the Low Luminance Deficit (LLD) Letter Score Categories in the Study Eye [Count of Participants; unit: Participants]
  <33 Letters | 236 | 235 | 471
  ≥33 Letters | 95 | 98 | 193
  Missing/Invalid | 3 | 4 | 7
Choroidal Neovascularization (CNV) Lesion Type in the Study Eye by Fundus Fluorescein Angiography [Count of Participants; unit: Participants]
  Occult | 177 | 174 | 351
  Classic | 84 | 73 | 157
  Minimally Classic | 32 | 30 | 62
  Retinal Angiomatous Proliferation (RAP) | 14 | 27 | 41
  Predominantly Classic | 17 | 19 | 36
  Polypoidal Choroidal Vasculopathy (PCV) | 6 | 6 | 12
  Missing | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in BCVA in the Study Eye Averaged Over Weeks 40, 44, and 48
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity. The Mixed Model of Repeated Measures (MMRM) analysis adjusted for treatment arm, visit, visit-by-treatment arm interaction, baseline BCVA (continuous), baseline BCVA (≥74, 73-55, and ≤54 letters), baseline LLD (<33 and ≥33 letters), and region (U.S. and Canada, Asia, and rest of the world). An unstructured covariance structure was used. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were implicitly imputed by MMRM. Invalid BCVA values were excluded from analysis. 95% CI is a rounding of 95.03% CI.
Time Frame: From Baseline through Week 48
Population: ITT Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization.
Measure: Mean (95% Confidence Interval); unit: ETDRS Letters
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 334 | 337
ETDRS Letters | 5.8 [4.6 to 7.1] | 5.1 [3.9 to 6.4]
Statistical Analysis 1: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; The null hypothesis, H0: μ(faricimab) - μ(aflibercept) ≤-4 letters; the alternative hypothesis, Ha: μ(faricimab) - μ(aflibercept) >-4 letters. A sample size of approximately 320 participants in each arm provided greater than 90% power to show non-inferiority of faricimab to aflibercept in the change from baseline BCVA averaged over Weeks 40, 44, and 48 in the ITT population, using a non-inferiority margin of 4 letters at the one-sided 0.02485 significance level; Test type: Non-Inferiority — If the lower bound of a two-sided 95.03% confidence interval (CI) for the difference in adjusted means of the two treatments (faricimab minus aflibercept) is greater than -4 letters (the non-inferiority margin), then faricimab is considered non-inferior to aflibercept; Adjusted mean difference = 0.7, 95% CI 2-sided [-1.1 to 2.5], Standard Error of Mean 0.91 — The treatment difference in adjusted means of change from baseline BCVA is the calculated difference of Arm A: Faricimab and Arm B: Aflibercept. MMRM adjustments are listed in the outcome measure description

2. Secondary Outcome: Change From Baseline in BCVA in the Study Eye Averaged Over Weeks 52, 56, and 60
Description: as for outcome 1
Time Frame: From Baseline through Week 60
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ETDRS Letters
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 334 | 337
ETDRS Letters | 5.4 [4.0 to 6.8] | 4.6 [3.3 to 6.0]
Statistical Analysis 1: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Treatment Difference in Adjusted Means at Weeks 52-60; Test type: Other; Adjusted mean difference = 0.7, 95% CI 2-sided [-1.2 to 2.7], Standard Error of Mean 0.99 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in BCVA in the Study Eye Over Time
Description: as for outcome 1
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, 100, 104, 108, and 112
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ETDRS Letters
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 334 | 337
ETDRS Letters
  Week 4 | 4.0 [3.2 to 4.8] | 3.6 [2.8 to 4.4]
  Week 8 | 5.5 [4.6 to 6.4] | 4.5 [3.6 to 5.4]
  Week 12 | 6.4 [5.5 to 7.4] | 5.3 [4.4 to 6.2]
  Week 16 | 6.8 [5.8 to 7.8] | 5.2 [4.2 to 6.2]
  Week 20 | 6.6 [5.5 to 7.6] | 4.9 [3.9 to 6.0]
  Week 24 | 6.4 [5.2 to 7.5] | 5.1 [4.0 to 6.3]
  Week 28 | 6.2 [5.1 to 7.3] | 5.6 [4.5 to 6.7]
  Week 32 | 6.2 [4.9 to 7.4] | 5.1 [3.8 to 6.3]
  Week 36 | 6.5 [5.3 to 7.7] | 5.5 [4.3 to 6.7]
  Week 40 | 6.1 [4.9 to 7.4] | 5.1 [3.9 to 6.4]
  Week 44 | 5.8 [4.5 to 7.1] | 5.1 [3.8 to 6.4]
  Week 48 | 5.5 [4.1 to 6.9] | 5.2 [3.8 to 6.5]
  Week 52 | 5.6 [4.2 to 7.1] | 4.5 [3.1 to 5.9]
  Week 56 | 5.5 [4.1 to 6.9] | 4.7 [3.3 to 6.1]
  Week 60 | 4.9 [3.5 to 6.3] | 4.7 [3.2 to 6.1]
  Week 64 | 5.5 [4.1 to 6.9] | 4.8 [3.5 to 6.2]
  Week 68 | 5.3 [3.9 to 6.8] | 4.6 [3.2 to 6.1]
  Week 72 | 4.8 [3.3 to 6.3] | 4.0 [2.5 to 5.4]
  Week 76 | 4.7 [3.1 to 6.2] | 4.4 [2.9 to 5.9]
  Week 80 | 4.6 [3.1 to 6.1] | 3.5 [2.0 to 5.1]
  Week 84 | 4.5 [3.0 to 6.1] | 3.5 [2.0 to 5.1]
  Week 88 | 4.3 [2.7 to 5.9] | 3.7 [2.1 to 5.2]
  Week 92 | 4.2 [2.6 to 5.9] | 3.7 [2.1 to 5.3]
  Week 96 | 4.2 [2.5 to 5.8] | 3.7 [2.0 to 5.3]
  Week 100 | 4.3 [2.7 to 5.9] | 3.6 [2.0 to 5.2]
  Week 104 | 4.1 [2.5 to 5.8] | 3.6 [2.0 to 5.2]
  Week 108 | 3.6 [1.8 to 5.3] | 3.2 [1.5 to 4.9]
  Week 112 | 3.5 [1.8 to 5.2] | 3.1 [1.4 to 4.8]

4. Secondary Outcome: Percentage of Participants Gaining Greater Than or Equal to (≥)15, ≥10, ≥5, or ≥0 Letters From the Baseline BCVA in the Study Eye Averaged Over Weeks 40, 44, and 48
Description: BCVA was measured on the ETDRS chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity. For each participant, an average BCVA value was calculated across the three visits, and this averaged value was used to determine if the endpoint was met. The results were summarized as the percentage of participants per treatment arm who met the endpoint. The weighted percentage of participants was based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥74 letters, 73-55 letters, and ≤54 letters), baseline LLD (≥33 letters and <33 letters), and region (U.S. and Canada vs. rest of the world). Treatment policy strategy and hypothetical strategy were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded. 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: Baseline, average of Weeks 40, 44, and 48
Population: ITT Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization. Participants with at least one non-missing, valid assessment at Weeks 40, 44, or 48 were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 292 | 300
Percentage of participants
  Gaining ≥15 Letters | 20.0 [15.6 to 24.4] | 15.7 [11.9 to 19.6]
  Gaining ≥10 Letters | 37.1 [31.7 to 42.4] | 31.7 [26.7 to 36.8]
  Gaining ≥5 Letters | 59.2 [53.7 to 64.7] | 58.0 [52.6 to 63.5]
  Gaining ≥0 Letters | 75.6 [70.8 to 80.3] | 76.8 [72.1 to 81.4]
Statistical Analysis 1: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Gaining ≥15 Letters: Treatment Difference at Weeks 40-48; Test type: Other; Difference in CMH Weighted Percentage = 4.3, 95% CI 2-sided [-1.6 to 10.1] — The treatment difference in CMH weighted percentage of participants gaining ≥15 letters is the calculated difference of Arm A: Faricimab and Arm B: Aflibercept
Statistical Analysis 2: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Gaining ≥10 Letters: Treatment Difference at Weeks 40-48; Test type: Other; Difference in CMH Weighted Percentage = 5.4, 95% CI 2-sided [-2.0 to 12.7] — The treatment difference in CMH weighted percentage of participants gaining ≥10 letters is the calculated difference of Arm A: Faricimab and Arm B: Aflibercept
Statistical Analysis 3: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Gaining ≥5 Letters: Treatment Difference at Weeks 40-48; Test type: Other; Difference in CMH Weighted Percentage = 1.2, 95% CI 2-sided [-6.6 to 8.9] — The treatment difference in CMH weighted percentage of participants gaining ≥5 letters is the calculated difference of Arm A: Faricimab and Arm B: Aflibercept
Statistical Analysis 4: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Gaining ≥0 Letters: Treatment Difference at Weeks 40-48; Test type: Other; Difference in CMH Weighted Percentage = -1.2, 95% CI 2-sided [-7.9 to 5.4] — The treatment difference in CMH weighted percentage of participants gaining ≥0 letters is the calculated difference of Arm A: Faricimab and Arm B: Aflibercept

5. Secondary Outcome: Percentage of Participants Gaining ≥15 Letters From the Baseline BCVA in the Study Eye Averaged Over Weeks 52, 56, and 60
Description: as for outcome 4
Time Frame: Baseline, average of Weeks 52, 56, and 60
Population: ITT Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization. Participants with at least one non-missing, valid assessment at Weeks 52, 56, or 60 were included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 277 | 283
Percentage of participants | 19.2 [15.0 to 23.5] | 16.6 [12.5 to 20.6]
Statistical Analysis 1: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Treatment Difference in CMH Weighted Percentages at Weeks 52-60; Test type: Other; Difference in CMH Weighted Percentage = 2.7, 95% CI 2-sided [-3.2 to 8.5] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Percentage of Participants Gaining ≥15 Letters From the Baseline BCVA in the Study Eye Over Time
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. The weighted percentage of participants was based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥74 letters, 73-55 letters, and ≤54 letters), baseline LLD (≥33 letters and <33 letters), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded from analysis. 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: as for outcome 3
Population: ITT Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization. At a given timepoint, the number analyzed includes participants with a non-missing, valid assessment at that timepoint.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 334 | 337
Percentage of participants
  Week 4: number analyzed (Participants) | 327 | 331
  Week 4 | 10.1 [6.9 to 13.2] | 6.3 [3.8 to 8.8]
  Week 8: number analyzed (Participants) | 325 | 325
  Week 8 | 13.7 [10.1 to 17.3] | 8.1 [5.3 to 10.9]
  Week 12: number analyzed (Participants) | 322 | 326
  Week 12 | 16.7 [12.8 to 20.5] | 10.1 [7.0 to 13.1]
  Week 16: number analyzed (Participants) | 322 | 320
  Week 16 | 17.7 [13.7 to 21.6] | 13.4 [10.0 to 16.9]
  Week 20: number analyzed (Participants) | 308 | 308
  Week 20 | 19.1 [14.9 to 23.2] | 12.7 [9.1 to 16.2]
  Week 24: number analyzed (Participants) | 278 | 285
  Week 24 | 22.1 [17.4 to 26.7] | 13.3 [9.6 to 17.0]
  Week 28: number analyzed (Participants) | 284 | 276
  Week 28 | 20.8 [16.4 to 25.2] | 16.2 [12.1 to 20.3]
  Week 32: number analyzed (Participants) | 293 | 285
  Week 32 | 21.6 [17.0 to 26.1] | 15.1 [11.3 to 18.9]
  Week 36: number analyzed (Participants) | 286 | 297
  Week 36 | 21.4 [16.8 to 26.0] | 15.7 [11.8 to 19.6]
  Week 40: number analyzed (Participants) | 287 | 291
  Week 40 | 22.1 [17.5 to 26.7] | 15.6 [11.7 to 19.5]
  Week 44: number analyzed (Participants) | 278 | 274
  Week 44 | 22.2 [17.5 to 26.8] | 17.4 [13.2 to 21.6]
  Week 48: number analyzed (Participants) | 273 | 279
  Week 48 | 21.2 [16.7 to 25.8] | 19.7 [15.3 to 24.0]
  Week 52: number analyzed (Participants) | 272 | 278
  Week 52 | 22.5 [17.8 to 27.2] | 18.3 [14.0 to 22.7]
  Week 56: number analyzed (Participants) | 273 | 279
  Week 56 | 23.1 [18.4 to 27.8] | 18.8 [14.6 to 23.0]
  Week 60: number analyzed (Participants) | 268 | 276
  Week 60 | 21.3 [16.7 to 25.9] | 17.4 [13.3 to 21.5]
  Week 64: number analyzed (Participants) | 253 | 276
  Week 64 | 20.3 [15.6 to 25.0] | 20.1 [15.7 to 24.6]
  Week 68: number analyzed (Participants) | 260 | 269
  Week 68 | 23.2 [18.3 to 28.1] | 18.5 [14.1 to 22.8]
  Week 72: number analyzed (Participants) | 262 | 274
  Week 72 | 21.1 [16.5 to 25.8] | 17.4 [13.1 to 21.6]
  Week 76: number analyzed (Participants) | 255 | 260
  Week 76 | 22.9 [18.0 to 27.8] | 18.0 [13.7 to 22.3]
  Week 80: number analyzed (Participants) | 254 | 268
  Week 80 | 19.7 [14.9 to 24.5] | 18.8 [14.4 to 23.2]
  Week 84: number analyzed (Participants) | 257 | 270
  Week 84 | 21.1 [16.4 to 25.9] | 18.3 [14.0 to 22.5]
  Week 88: number analyzed (Participants) | 256 | 267
  Week 88 | 24.6 [19.7 to 29.6] | 18.6 [14.3 to 23.0]
  Week 92: number analyzed (Participants) | 247 | 266
  Week 92 | 21.4 [16.5 to 26.3] | 19.5 [14.9 to 24.0]
  Week 96: number analyzed (Participants) | 249 | 258
  Week 96 | 23.0 [18.1 to 27.9] | 20.2 [15.7 to 24.6]
  Week 100: number analyzed (Participants) | 248 | 258
  Week 100 | 21.5 [16.7 to 26.3] | 18.2 [13.9 to 22.5]
  Week 104: number analyzed (Participants) | 250 | 263
  Week 104 | 22.9 [17.9 to 27.8] | 18.6 [14.2 to 22.9]
  Week 108: number analyzed (Participants) | 246 | 256
  Week 108 | 21.9 [17.0 to 26.7] | 19.0 [14.6 to 23.4]
  Week 112: number analyzed (Participants) | 247 | 259
  Week 112 | 24.0 [19.1 to 29.0] | 19.2 [14.6 to 23.7]

7. Secondary Outcome: Percentage of Participants Gaining ≥10 Letters From the Baseline BCVA in the Study Eye Over Time
Description: as for outcome 6
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 334 | 337
Percentage of participants
  Week 4: number analyzed (Participants) | 327 | 331
  Week 4 | 20.1 [16.0 to 24.2] | 16.0 [12.3 to 19.7]
  Week 8: number analyzed (Participants) | 325 | 325
  Week 8 | 28.6 [23.9 to 33.3] | 25.3 [20.9 to 29.8]
  Week 12: number analyzed (Participants) | 322 | 326
  Week 12 | 31.4 [26.5 to 36.3] | 30.3 [25.5 to 35.1]
  Week 16: number analyzed (Participants) | 322 | 320
  Week 16 | 36.9 [31.8 to 41.9] | 31.9 [27.0 to 36.7]
  Week 20: number analyzed (Participants) | 308 | 308
  Week 20 | 39.1 [34.0 to 44.2] | 30.3 [25.4 to 35.2]
  Week 24: number analyzed (Participants) | 278 | 285
  Week 24 | 41.4 [36.0 to 46.9] | 34.0 [28.7 to 39.3]
  Week 28: number analyzed (Participants) | 284 | 276
  Week 28 | 38.9 [33.5 to 44.3] | 34.8 [29.5 to 40.1]
  Week 32: number analyzed (Participants) | 293 | 285
  Week 32 | 38.6 [33.2 to 44.0] | 32.4 [27.2 to 37.7]
  Week 36: number analyzed (Participants) | 286 | 297
  Week 36 | 37.1 [31.6 to 42.6] | 34.0 [28.8 to 39.2]
  Week 40: number analyzed (Participants) | 287 | 291
  Week 40 | 36.9 [31.5 to 42.3] | 33.9 [28.6 to 39.2]
  Week 44: number analyzed (Participants) | 278 | 274
  Week 44 | 39.5 [33.9 to 45.0] | 34.3 [29.0 to 39.7]
  Week 48: number analyzed (Participants) | 273 | 279
  Week 48 | 36.8 [31.3 to 42.3] | 36.8 [31.4 to 42.2]
  Week 52: number analyzed (Participants) | 272 | 278
  Week 52 | 38.7 [33.2 to 44.2] | 37.7 [32.2 to 43.2]
  Week 56: number analyzed (Participants) | 273 | 279
  Week 56 | 40.3 [34.8 to 45.8] | 36.2 [30.8 to 41.6]
  Week 60: number analyzed (Participants) | 268 | 276
  Week 60 | 40.1 [34.7 to 45.5] | 34.8 [29.4 to 40.3]
  Week 64: number analyzed (Participants) | 253 | 276
  Week 64 | 37.2 [31.4 to 43.0] | 36.6 [31.1 to 42.0]
  Week 68: number analyzed (Participants) | 260 | 269
  Week 68 | 40.0 [34.3 to 45.7] | 33.3 [27.8 to 38.7]
  Week 72: number analyzed (Participants) | 262 | 274
  Week 72 | 40.1 [34.4 to 45.8] | 34.3 [28.8 to 39.8]
  Week 76: number analyzed (Participants) | 255 | 260
  Week 76 | 39.4 [33.7 to 45.2] | 33.5 [28.0 to 39.0]
  Week 80: number analyzed (Participants) | 254 | 268
  Week 80 | 35.5 [29.8 to 41.2] | 33.0 [27.7 to 38.4]
  Week 84: number analyzed (Participants) | 257 | 270
  Week 84 | 38.2 [32.5 to 43.9] | 34.3 [28.9 to 39.7]
  Week 88: number analyzed (Participants) | 256 | 267
  Week 88 | 38.9 [33.2 to 44.7] | 33.6 [28.3 to 39.0]
  Week 92: number analyzed (Participants) | 247 | 266
  Week 92 | 37.8 [31.9 to 43.7] | 35.3 [29.7 to 40.8]
  Week 96: number analyzed (Participants) | 249 | 258
  Week 96 | 39.6 [33.7 to 45.4] | 35.8 [30.3 to 41.4]
  Week 100: number analyzed (Participants) | 248 | 258
  Week 100 | 38.5 [32.7 to 44.4] | 36.4 [30.8 to 42.0]
  Week 104: number analyzed (Participants) | 250 | 263
  Week 104 | 38.7 [32.9 to 44.6] | 38.9 [33.3 to 44.5]
  Week 108: number analyzed (Participants) | 246 | 256
  Week 108 | 35.1 [29.3 to 40.9] | 36.6 [30.9 to 42.2]
  Week 112: number analyzed (Participants) | 247 | 259
  Week 112 | 39.5 [33.8 to 45.3] | 34.9 [29.3 to 40.5]

8. Secondary Outcome: Percentage of Participants Gaining ≥5 Letters From the Baseline BCVA in the Study Eye Over Time
Description: as for outcome 6
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 334 | 337
Percentage of participants
  Week 4: number analyzed (Participants) | 327 | 331
  Week 4 | 47.6 [42.3 to 52.8] | 45.6 [40.4 to 50.9]
  Week 8: number analyzed (Participants) | 325 | 325
  Week 8 | 57.8 [52.5 to 63.0] | 52.3 [47.2 to 57.5]
  Week 12: number analyzed (Participants) | 322 | 326
  Week 12 | 61.5 [56.3 to 66.8] | 55.0 [49.7 to 60.2]
  Week 16: number analyzed (Participants) | 322 | 320
  Week 16 | 61.8 [56.5 to 67.0] | 54.0 [48.7 to 59.3]
  Week 20: number analyzed (Participants) | 308 | 308
  Week 20 | 60.2 [54.8 to 65.6] | 55.5 [50.0 to 60.9]
  Week 24: number analyzed (Participants) | 278 | 285
  Week 24 | 63.4 [57.9 to 68.9] | 53.6 [48.0 to 59.3]
  Week 28: number analyzed (Participants) | 284 | 276
  Week 28 | 60.8 [55.3 to 66.3] | 61.4 [55.8 to 67.0]
  Week 32: number analyzed (Participants) | 293 | 285
  Week 32 | 60.5 [55.1 to 65.9] | 56.4 [50.8 to 62.0]
  Week 36: number analyzed (Participants) | 286 | 297
  Week 36 | 60.5 [55.0 to 66.0] | 58.5 [53.0 to 64.0]
  Week 40: number analyzed (Participants) | 287 | 291
  Week 40 | 59.1 [53.6 to 64.6] | 54.5 [48.9 to 60.2]
  Week 44: number analyzed (Participants) | 278 | 274
  Week 44 | 60.3 [54.7 to 65.9] | 59.0 [53.3 to 64.6]
  Week 48: number analyzed (Participants) | 273 | 279
  Week 48 | 59.3 [53.7 to 65.0] | 58.8 [53.2 to 64.4]
  Week 52: number analyzed (Participants) | 272 | 278
  Week 52 | 62.6 [57.0 to 68.1] | 58.5 [52.8 to 64.1]
  Week 56: number analyzed (Participants) | 273 | 279
  Week 56 | 58.6 [53.0 to 64.2] | 54.4 [48.7 to 60.2]
  Week 60: number analyzed (Participants) | 268 | 276
  Week 60 | 60.4 [54.8 to 66.0] | 57.4 [51.6 to 63.1]
  Week 64: number analyzed (Participants) | 253 | 276
  Week 64 | 59.3 [53.5 to 65.2] | 55.1 [49.3 to 60.9]
  Week 68: number analyzed (Participants) | 260 | 269
  Week 68 | 60.4 [54.7 to 66.1] | 57.0 [51.2 to 62.7]
  Week 72: number analyzed (Participants) | 262 | 274
  Week 72 | 59.8 [54.0 to 65.5] | 52.3 [46.5 to 58.1]
  Week 76: number analyzed (Participants) | 255 | 260
  Week 76 | 59.3 [53.5 to 65.1] | 55.0 [49.1 to 60.9]
  Week 80: number analyzed (Participants) | 254 | 268
  Week 80 | 55.2 [49.3 to 61.2] | 55.5 [49.6 to 61.3]
  Week 84: number analyzed (Participants) | 257 | 270
  Week 84 | 58.4 [52.6 to 64.2] | 55.6 [49.8 to 61.4]
  Week 88: number analyzed (Participants) | 256 | 267
  Week 88 | 59.3 [53.5 to 65.1] | 53.8 [48.0 to 59.6]
  Week 92: number analyzed (Participants) | 247 | 266
  Week 92 | 56.8 [50.8 to 62.9] | 56.0 [50.3 to 61.8]
  Week 96: number analyzed (Participants) | 249 | 258
  Week 96 | 58.2 [52.2 to 64.1] | 57.5 [51.7 to 63.4]
  Week 100: number analyzed (Participants) | 248 | 258
  Week 100 | 59.1 [53.2 to 65.1] | 57.1 [51.2 to 63.0]
  Week 104: number analyzed (Participants) | 250 | 263
  Week 104 | 59.8 [54.0 to 65.7] | 54.8 [48.9 to 60.7]
  Week 108: number analyzed (Participants) | 246 | 256
  Week 108 | 53.6 [47.7 to 59.6] | 54.1 [48.2 to 60.1]
  Week 112: number analyzed (Participants) | 247 | 259
  Week 112 | 57.3 [51.4 to 63.2] | 53.5 [47.6 to 59.5]

9. Secondary Outcome: Percentage of Participants Gaining ≥0 Letters From the Baseline BCVA in the Study Eye Over Time
Description: as for outcome 6
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 334 | 337
Percentage of participants
  Week 4: number analyzed (Participants) | 327 | 331
  Week 4 | 78.9 [74.5 to 83.2] | 77.6 [73.3 to 81.9]
  Week 8: number analyzed (Participants) | 325 | 325
  Week 8 | 80.7 [76.4 to 84.9] | 78.3 [73.9 to 82.7]
  Week 12: number analyzed (Participants) | 322 | 326
  Week 12 | 84.2 [80.3 to 88.1] | 81.4 [77.3 to 85.6]
  Week 16: number analyzed (Participants) | 322 | 320
  Week 16 | 84.8 [80.9 to 88.7] | 78.8 [74.6 to 83.1]
  Week 20: number analyzed (Participants) | 308 | 308
  Week 20 | 80.8 [76.5 to 85.2] | 79.6 [75.2 to 83.9]
  Week 24: number analyzed (Participants) | 278 | 285
  Week 24 | 81.9 [77.5 to 86.3] | 79.6 [75.1 to 84.1]
  Week 28: number analyzed (Participants) | 284 | 276
  Week 28 | 77.8 [73.1 to 82.6] | 82.3 [77.9 to 86.7]
  Week 32: number analyzed (Participants) | 293 | 285
  Week 32 | 78.7 [74.2 to 83.1] | 76.3 [71.5 to 81.0]
  Week 36: number analyzed (Participants) | 286 | 297
  Week 36 | 78.9 [74.3 to 83.5] | 81.0 [76.6 to 85.4]
  Week 40: number analyzed (Participants) | 287 | 291
  Week 40 | 77.1 [72.5 to 81.7] | 80.7 [76.3 to 85.2]
  Week 44: number analyzed (Participants) | 278 | 274
  Week 44 | 77.0 [72.3 to 81.7] | 78.3 [73.6 to 83.0]
  Week 48: number analyzed (Participants) | 273 | 279
  Week 48 | 77.0 [72.2 to 81.8] | 76.4 [71.5 to 81.3]
  Week 52: number analyzed (Participants) | 272 | 278
  Week 52 | 77.4 [72.6 to 82.2] | 75.7 [70.7 to 80.6]
  Week 56: number analyzed (Participants) | 273 | 279
  Week 56 | 76.3 [71.4 to 81.1] | 78.7 [73.9 to 83.5]
  Week 60: number analyzed (Participants) | 268 | 276
  Week 60 | 74.4 [69.3 to 79.5] | 77.5 [72.6 to 82.3]
  Week 64: number analyzed (Participants) | 253 | 276
  Week 64 | 77.7 [72.8 to 82.6] | 73.7 [68.6 to 78.8]
  Week 68: number analyzed (Participants) | 260 | 269
  Week 68 | 74.9 [69.8 to 80.0] | 77.7 [72.8 to 82.6]
  Week 72: number analyzed (Participants) | 262 | 274
  Week 72 | 74.9 [69.9 to 79.8] | 74.8 [69.8 to 79.8]
  Week 76: number analyzed (Participants) | 255 | 260
  Week 76 | 75.7 [70.8 to 80.7] | 72.0 [66.6 to 77.4]
  Week 80: number analyzed (Participants) | 254 | 268
  Week 80 | 75.5 [70.4 to 80.5] | 74.4 [69.3 to 79.5]
  Week 84: number analyzed (Participants) | 257 | 270
  Week 84 | 75.5 [70.5 to 80.5] | 72.5 [67.3 to 77.7]
  Week 88: number analyzed (Participants) | 256 | 267
  Week 88 | 74.8 [69.6 to 80.0] | 71.7 [66.4 to 76.9]
  Week 92: number analyzed (Participants) | 247 | 266
  Week 92 | 75.0 [69.9 to 80.2] | 70.6 [65.3 to 75.9]
  Week 96: number analyzed (Participants) | 249 | 258
  Week 96 | 74.7 [69.6 to 79.9] | 71.1 [65.7 to 76.5]
  Week 100: number analyzed (Participants) | 248 | 258
  Week 100 | 74.6 [69.4 to 79.8] | 69.7 [64.2 to 75.2]
  Week 104: number analyzed (Participants) | 250 | 263
  Week 104 | 73.8 [68.6 to 79.1] | 71.2 [66.0 to 76.5]
  Week 108: number analyzed (Participants) | 246 | 256
  Week 108 | 73.4 [68.2 to 78.7] | 73.7 [68.4 to 79.0]
  Week 112: number analyzed (Participants) | 247 | 259
  Week 112 | 72.8 [67.5 to 78.1] | 70.9 [65.5 to 76.3]

10. Secondary Outcome: Percentage of Participants Avoiding a Loss of ≥15, ≥10, or ≥5 Letters From the Baseline BCVA in the Study Eye Averaged Over Weeks 40, 44, and 48
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. For each participant, an average BCVA value was calculated across the three visits, and this averaged value was then used to determine if the endpoint was met. The results were summarized as the percentage of participants per treatment arm who met the endpoint. The weighted percentage of participants was based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥74 letters, 73-55 letters, and ≤54 letters), baseline LLD (≥33 letters and <33 letters), and region (U.S. and Canada vs. rest of the world). Treatment policy strategy and hypothetical strategy were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded. 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: Baseline, average of Weeks 40, 44, and 48
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 292 | 300
Percentage of participants
  Avoiding a Loss of ≥15 Letters | 95.4 [93.0 to 97.7] | 94.1 [91.5 to 96.7]
  Avoiding a Loss of ≥10 Letters | 91.6 [88.6 to 94.7] | 92.0 [89.1 to 95.0]
  Avoiding a Loss of ≥5 Letters | 88.0 [84.3 to 91.6] | 86.8 [83.0 to 90.5]
Statistical Analysis 1: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Avoiding a Loss of ≥15 Letters: Treatment Difference at Weeks 40-48; Test type: Other; Difference in CMH Weighted Percentage = 1.3, 95% CI 2-sided [-2.2 to 4.8] — The treatment difference in CMH weighted percentage of participants avoiding a loss of ≥15 letters is the calculated difference of Arm A: Faricimab and Arm B: Aflibercept
Statistical Analysis 2: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Avoiding a Loss of ≥10 Letters: Treatment Difference at Weeks 40-48; Test type: Other; Difference in CMH Weighted Percentage = -0.4, 95% CI 2-sided [-4.6 to 3.9] — The treatment difference in CMH weighted percentage of participants avoiding a loss of ≥10 letters is the calculated difference of Arm A: Faricimab and Arm B: Aflibercept
Statistical Analysis 3: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Avoiding a Loss of ≥5 Letters: Treatment Difference at Weeks 40-48; Test type: Other; Difference in CMH Weighted Percentage = 1.2, 95% CI 2-sided [-4.0 to 6.4] — The treatment difference in CMH weighted percentage of participants avoiding a loss of ≥5 letters is the calculated difference of Arm A: Faricimab and Arm B: Aflibercept

11. Secondary Outcome: Percentage of Participants Avoiding a Loss of ≥15 Letters From the Baseline BCVA in the Study Eye Averaged Over Weeks 52, 56, and 60
Description: as for outcome 10
Time Frame: Baseline, average of Weeks 52, 56, and 60
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 277 | 283
Percentage of participants | 93.9 [91.3 to 96.5] | 94.1 [91.4 to 96.8]
Statistical Analysis 1: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Treatment Difference in CMH Weighted Percentages at Weeks 52-60; Test type: Other; Difference in CMH Weighted Percentage = -0.2, 95% CI 2-sided [-3.9 to 3.6] — [estimate comment as in outcome 10, analysis 1]

12. Secondary Outcome: Percentage of Participants Avoiding a Loss of ≥15 Letters From the Baseline BCVA in the Study Eye Over Time
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The weighted percentage of participants avoiding a loss of letters in BCVA from baseline was based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥74 letters, 73-55 letters, and ≤54 letters), baseline LLD (≥33 letters and <33 letters), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded from analysis. 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 334 | 337
Percentage of participants
  Week 4: number analyzed (Participants) | 327 | 331
  Week 4 | 97.6 [95.9 to 99.2] | 99.0 [98.0 to 100.0]
  Week 8: number analyzed (Participants) | 325 | 325
  Week 8 | 97.6 [96.0 to 99.2] | 98.7 [97.6 to 99.9]
  Week 12: number analyzed (Participants) | 322 | 326
  Week 12 | 98.2 [96.7 to 99.6] | 97.5 [95.8 to 99.1]
  Week 16: number analyzed (Participants) | 322 | 320
  Week 16 | 98.1 [96.7 to 99.6] | 97.0 [95.3 to 98.8]
  Week 20: number analyzed (Participants) | 308 | 308
  Week 20 | 97.4 [95.7 to 99.1] | 94.9 [92.5 to 97.3]
  Week 24: number analyzed (Participants) | 278 | 285
  Week 24 | 97.2 [95.3 to 99.1] | 97.5 [95.8 to 99.3]
  Week 28: number analyzed (Participants) | 284 | 276
  Week 28 | 95.9 [93.8 to 98.1] | 96.7 [94.6 to 98.8]
  Week 32: number analyzed (Participants) | 293 | 285
  Week 32 | 95.4 [93.1 to 97.7] | 95.7 [93.5 to 98.0]
  Week 36: number analyzed (Participants) | 286 | 297
  Week 36 | 95.2 [92.8 to 97.6] | 95.4 [93.1 to 97.7]
  Week 40: number analyzed (Participants) | 287 | 291
  Week 40 | 96.6 [94.5 to 98.6] | 94.2 [91.6 to 96.8]
  Week 44: number analyzed (Participants) | 278 | 274
  Week 44 | 95.7 [93.5 to 98.0] | 93.9 [91.2 to 96.6]
  Week 48: number analyzed (Participants) | 273 | 279
  Week 48 | 94.0 [91.3 to 96.7] | 93.3 [90.4 to 96.1]
  Week 52: number analyzed (Participants) | 272 | 278
  Week 52 | 93.5 [90.8 to 96.2] | 93.5 [90.7 to 96.3]
  Week 56: number analyzed (Participants) | 273 | 279
  Week 56 | 94.7 [92.2 to 97.2] | 95.0 [92.5 to 97.5]
  Week 60: number analyzed (Participants) | 268 | 276
  Week 60 | 93.6 [90.8 to 96.4] | 92.6 [89.7 to 95.6]
  Week 64: number analyzed (Participants) | 253 | 276
  Week 64 | 94.1 [91.3 to 96.9] | 92.9 [89.9 to 95.9]
  Week 68: number analyzed (Participants) | 260 | 269
  Week 68 | 92.6 [89.6 to 95.6] | 92.9 [89.9 to 95.8]
  Week 72: number analyzed (Participants) | 262 | 274
  Week 72 | 93.5 [90.7 to 96.3] | 91.3 [88.2 to 94.4]
  Week 76: number analyzed (Participants) | 255 | 260
  Week 76 | 94.2 [91.6 to 96.8] | 92.7 [89.8 to 95.7]
  Week 80: number analyzed (Participants) | 254 | 268
  Week 80 | 93.6 [90.9 to 96.4] | 90.7 [87.4 to 93.9]
  Week 84: number analyzed (Participants) | 257 | 270
  Week 84 | 92.8 [89.9 to 95.7] | 91.5 [88.4 to 94.5]
  Week 88: number analyzed (Participants) | 256 | 267
  Week 88 | 93.1 [90.3 to 96.0] | 90.4 [87.2 to 93.7]
  Week 92: number analyzed (Participants) | 247 | 266
  Week 92 | 92.1 [89.1 to 95.2] | 93.2 [90.5 to 95.9]
  Week 96: number analyzed (Participants) | 249 | 258
  Week 96 | 91.6 [88.4 to 94.8] | 88.9 [85.3 to 92.5]
  Week 100: number analyzed (Participants) | 248 | 258
  Week 100 | 92.7 [89.8 to 95.6] | 89.5 [86.0 to 93.0]
  Week 104: number analyzed (Participants) | 250 | 263
  Week 104 | 93.2 [90.3 to 96.1] | 90.7 [87.4 to 93.9]
  Week 108: number analyzed (Participants) | 246 | 256
  Week 108 | 92.0 [88.9 to 95.1] | 89.6 [86.0 to 93.2]
  Week 112: number analyzed (Participants) | 247 | 259
  Week 112 | 90.6 [87.3 to 93.9] | 88.8 [85.1 to 92.4]

13. Secondary Outcome: Percentage of Participants Avoiding a Loss of ≥10 Letters From the Baseline BCVA in the Study Eye Over Time
Description: as for outcome 12
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 334 | 337
Percentage of participants
  Week 4: number analyzed (Participants) | 327 | 331
  Week 4 | 95.1 [92.9 to 97.4] | 96.2 [94.3 to 98.2]
  Week 8: number analyzed (Participants) | 325 | 325
  Week 8 | 96.0 [94.0 to 98.0] | 96.9 [95.1 to 98.7]
  Week 12: number analyzed (Participants) | 322 | 326
  Week 12 | 96.3 [94.4 to 98.3] | 95.5 [93.3 to 97.7]
  Week 16: number analyzed (Participants) | 322 | 320
  Week 16 | 95.1 [92.8 to 97.4] | 92.6 [89.9 to 95.4]
  Week 20: number analyzed (Participants) | 308 | 308
  Week 20 | 93.9 [91.3 to 96.5] | 92.7 [89.9 to 95.4]
  Week 24: number analyzed (Participants) | 278 | 285
  Week 24 | 94.3 [91.7 to 96.9] | 94.4 [91.9 to 96.9]
  Week 28: number analyzed (Participants) | 284 | 276
  Week 28 | 93.5 [90.8 to 96.2] | 94.9 [92.3 to 97.4]
  Week 32: number analyzed (Participants) | 293 | 285
  Week 32 | 92.5 [89.6 to 95.3] | 92.9 [89.9 to 95.8]
  Week 36: number analyzed (Participants) | 286 | 297
  Week 36 | 93.2 [90.3 to 96.0] | 91.7 [88.6 to 94.7]
  Week 40: number analyzed (Participants) | 287 | 291
  Week 40 | 92.2 [89.2 to 95.2] | 91.8 [88.8 to 94.8]
  Week 44: number analyzed (Participants) | 278 | 274
  Week 44 | 92.3 [89.4 to 95.3] | 90.9 [87.7 to 94.2]
  Week 48: number analyzed (Participants) | 273 | 279
  Week 48 | 91.5 [88.3 to 94.6] | 91.5 [88.3 to 94.7]
  Week 52: number analyzed (Participants) | 272 | 278
  Week 52 | 91.7 [88.6 to 94.7] | 91.1 [87.8 to 94.4]
  Week 56: number analyzed (Participants) | 273 | 279
  Week 56 | 92.3 [89.3 to 95.3] | 90.4 [87.0 to 93.8]
  Week 60: number analyzed (Participants) | 268 | 276
  Week 60 | 90.7 [87.5 to 94.0] | 88.5 [85.0 to 92.1]
  Week 64: number analyzed (Participants) | 253 | 276
  Week 64 | 91.3 [88.0 to 94.6] | 90.3 [87.0 to 93.7]
  Week 68: number analyzed (Participants) | 260 | 269
  Week 68 | 92.2 [89.2 to 95.3] | 90.3 [86.9 to 93.7]
  Week 72: number analyzed (Participants) | 262 | 274
  Week 72 | 89.6 [86.2 to 93.1] | 88.1 [84.6 to 91.7]
  Week 76: number analyzed (Participants) | 255 | 260
  Week 76 | 89.2 [85.6 to 92.7] | 88.0 [84.3 to 91.8]
  Week 80: number analyzed (Participants) | 254 | 268
  Week 80 | 89.3 [85.7 to 92.9] | 86.4 [82.6 to 90.2]
  Week 84: number analyzed (Participants) | 257 | 270
  Week 84 | 89.0 [85.5 to 92.5] | 86.9 [83.2 to 90.7]
  Week 88: number analyzed (Participants) | 256 | 267
  Week 88 | 89.2 [85.7 to 92.7] | 85.2 [81.2 to 89.3]
  Week 92: number analyzed (Participants) | 247 | 266
  Week 92 | 87.7 [83.8 to 91.6] | 86.3 [82.4 to 90.1]
  Week 96: number analyzed (Participants) | 249 | 258
  Week 96 | 87.8 [84.0 to 91.5] | 85.7 [81.6 to 89.8]
  Week 100: number analyzed (Participants) | 248 | 258
  Week 100 | 88.6 [84.9 to 92.3] | 86.1 [82.1 to 90.1]
  Week 104: number analyzed (Participants) | 250 | 263
  Week 104 | 87.6 [83.7 to 91.5] | 85.3 [81.3 to 89.4]
  Week 108: number analyzed (Participants) | 246 | 256
  Week 108 | 85.2 [81.1 to 89.4] | 87.3 [83.4 to 91.2]
  Week 112: number analyzed (Participants) | 247 | 259
  Week 112 | 84.7 [80.5 to 88.9] | 84.2 [79.9 to 88.5]

14. Secondary Outcome: Percentage of Participants Avoiding a Loss of ≥5 Letters From the Baseline BCVA in the Study Eye Over Time
Description: as for outcome 12
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 334 | 337
Percentage of participants
  Week 4: number analyzed (Participants) | 327 | 331
  Week 4 | 90.5 [87.4 to 93.6] | 90.6 [87.5 to 93.6]
  Week 8: number analyzed (Participants) | 325 | 325
  Week 8 | 92.3 [89.6 to 95.1] | 90.6 [87.5 to 93.7]
  Week 12: number analyzed (Participants) | 322 | 326
  Week 12 | 92.2 [89.4 to 95.1] | 88.8 [85.4 to 92.1]
  Week 16: number analyzed (Participants) | 322 | 320
  Week 16 | 90.4 [87.3 to 93.6] | 87.4 [83.8 to 90.9]
  Week 20: number analyzed (Participants) | 308 | 308
  Week 20 | 89.3 [85.9 to 92.7] | 87.1 [83.5 to 90.7]
  Week 24: number analyzed (Participants) | 278 | 285
  Week 24 | 89.1 [85.6 to 92.6] | 88.8 [85.3 to 92.3]
  Week 28: number analyzed (Participants) | 284 | 276
  Week 28 | 88.2 [84.6 to 91.9] | 90.2 [86.7 to 93.6]
  Week 32: number analyzed (Participants) | 293 | 285
  Week 32 | 87.0 [83.3 to 90.7] | 85.8 [81.9 to 89.6]
  Week 36: number analyzed (Participants) | 286 | 297
  Week 36 | 88.3 [84.7 to 91.9] | 86.7 [82.9 to 90.4]
  Week 40: number analyzed (Participants) | 287 | 291
  Week 40 | 86.8 [83.1 to 90.6] | 87.4 [83.7 to 91.1]
  Week 44: number analyzed (Participants) | 278 | 274
  Week 44 | 85.2 [81.3 to 89.2] | 85.3 [81.2 to 89.4]
  Week 48: number analyzed (Participants) | 273 | 279
  Week 48 | 85.6 [81.6 to 89.6] | 83.5 [79.3 to 87.7]
  Week 52: number analyzed (Participants) | 272 | 278
  Week 52 | 84.8 [80.7 to 88.9] | 85.5 [81.4 to 89.6]
  Week 56: number analyzed (Participants) | 273 | 279
  Week 56 | 84.4 [80.4 to 88.5] | 83.7 [79.4 to 88.0]
  Week 60: number analyzed (Participants) | 268 | 276
  Week 60 | 81.5 [77.0 to 85.9] | 84.5 [80.4 to 88.6]
  Week 64: number analyzed (Participants) | 253 | 276
  Week 64 | 87.8 [84.0 to 91.7] | 85.3 [81.3 to 89.4]
  Week 68: number analyzed (Participants) | 260 | 269
  Week 68 | 85.0 [80.9 to 89.1] | 87.0 [83.1 to 90.9]
  Week 72: number analyzed (Participants) | 262 | 274
  Week 72 | 84.2 [80.0 to 88.3] | 81.1 [76.6 to 85.6]
  Week 76: number analyzed (Participants) | 255 | 260
  Week 76 | 83.5 [79.1 to 87.8] | 83.3 [78.9 to 87.7]
  Week 80: number analyzed (Participants) | 254 | 268
  Week 80 | 81.0 [76.3 to 85.6] | 81.9 [77.5 to 86.4]
  Week 84: number analyzed (Participants) | 257 | 270
  Week 84 | 82.6 [78.2 to 86.9] | 81.8 [77.4 to 86.3]
  Week 88: number analyzed (Participants) | 256 | 267
  Week 88 | 80.8 [76.2 to 85.4] | 78.8 [74.1 to 83.6]
  Week 92: number analyzed (Participants) | 247 | 266
  Week 92 | 81.7 [77.1 to 86.3] | 79.2 [74.5 to 83.9]
  Week 96: number analyzed (Participants) | 249 | 258
  Week 96 | 82.1 [77.6 to 86.6] | 78.1 [73.2 to 83.0]
  Week 100: number analyzed (Participants) | 248 | 258
  Week 100 | 81.7 [77.1 to 86.3] | 80.1 [75.4 to 84.8]
  Week 104: number analyzed (Participants) | 250 | 263
  Week 104 | 79.6 [74.7 to 84.4] | 80.5 [75.8 to 85.1]
  Week 108: number analyzed (Participants) | 246 | 256
  Week 108 | 79.7 [74.9 to 84.4] | 80.7 [75.9 to 85.4]
  Week 112: number analyzed (Participants) | 247 | 259
  Week 112 | 78.6 [73.7 to 83.4] | 78.9 [74.1 to 83.7]

15. Secondary Outcome: Percentage of Participants Gaining ≥15 Letters From the Baseline BCVA or Achieving BCVA Snellen Equivalent of 20/20 or Better (BCVA ≥84 Letters) in the Study Eye Averaged Over Weeks 40, 44, and 48
Description: as for outcome 4
Time Frame: Baseline, average of Weeks 40, 44, and 48
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 292 | 300
Percentage of participants | 24.3 [19.5 to 29.1] | 21.3 [16.8 to 25.7]
Statistical Analysis 1: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Treatment Difference in CMH Weighted Percentages at Weeks 40-48; Test type: Other; Difference in CMH Weighted Percentage = 3.0, 95% CI 2-sided [-3.6 to 9.5] — The treatment difference in CMH weighted percentage of participants gaining ≥15 letters or achieving BCVA ≥84 letters is the calculated difference of Arm A: Faricimab and Arm B: Aflibercept

16. Secondary Outcome: Percentage of Participants Gaining ≥15 Letters From the Baseline BCVA or Achieving BCVA Snellen Equivalent of 20/20 or Better (BCVA ≥84 Letters) in the Study Eye Over Time
Description: as for outcome 6
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 334 | 337
Percentage of participants
  Week 4: number analyzed (Participants) | 327 | 331
  Week 4 | 11.0 [7.7 to 14.3] | 8.1 [5.3 to 10.9]
  Week 8: number analyzed (Participants) | 325 | 325
  Week 8 | 16.3 [12.3 to 20.2] | 11.1 [7.8 to 14.4]
  Week 12: number analyzed (Participants) | 322 | 326
  Week 12 | 20.4 [16.2 to 24.7] | 14.9 [11.2 to 18.6]
  Week 16: number analyzed (Participants) | 322 | 320
  Week 16 | 20.5 [16.3 to 24.8] | 17.3 [13.4 to 21.3]
  Week 20: number analyzed (Participants) | 308 | 308
  Week 20 | 22.4 [17.9 to 26.9] | 17.7 [13.5 to 21.8]
  Week 24: number analyzed (Participants) | 278 | 285
  Week 24 | 25.5 [20.5 to 30.5] | 19.1 [14.7 to 23.4]
  Week 28: number analyzed (Participants) | 284 | 276
  Week 28 | 25.7 [20.8 to 30.5] | 20.0 [15.5 to 24.5]
  Week 32: number analyzed (Participants) | 293 | 285
  Week 32 | 27.3 [22.4 to 32.3] | 21.9 [17.3 to 26.5]
  Week 36: number analyzed (Participants) | 286 | 297
  Week 36 | 27.2 [22.1 to 32.2] | 23.7 [19.0 to 28.4]
  Week 40: number analyzed (Participants) | 287 | 291
  Week 40 | 26.0 [21.0 to 30.9] | 21.4 [16.8 to 25.9]
  Week 44: number analyzed (Participants) | 278 | 274
  Week 44 | 26.5 [21.5 to 31.6] | 22.8 [18.1 to 27.5]
  Week 48: number analyzed (Participants) | 273 | 279
  Week 48 | 24.9 [20.0 to 29.8] | 27.6 [22.5 to 32.6]
  Week 52: number analyzed (Participants) | 272 | 278
  Week 52 | 25.0 [20.1 to 30.0] | 23.8 [19.0 to 28.7]
  Week 56: number analyzed (Participants) | 273 | 279
  Week 56 | 26.4 [21.4 to 31.5] | 24.4 [19.7 to 29.1]
  Week 60: number analyzed (Participants) | 268 | 276
  Week 60 | 25.2 [20.2 to 30.2] | 22.7 [18.1 to 27.4]
  Week 64: number analyzed (Participants) | 253 | 276
  Week 64 | 24.2 [19.1 to 29.3] | 25.6 [20.6 to 30.5]
  Week 68: number analyzed (Participants) | 260 | 269
  Week 68 | 27.5 [22.2 to 32.8] | 24.3 [19.4 to 29.2]
  Week 72: number analyzed (Participants) | 262 | 274
  Week 72 | 26.1 [21.0 to 31.2] | 24.2 [19.4 to 29.0]
  Week 76: number analyzed (Participants) | 255 | 260
  Week 76 | 27.6 [22.2 to 32.9] | 23.6 [18.8 to 28.5]
  Week 80: number analyzed (Participants) | 254 | 268
  Week 80 | 24.1 [18.9 to 29.3] | 25.9 [20.9 to 31.0]
  Week 84: number analyzed (Participants) | 257 | 270
  Week 84 | 26.2 [21.0 to 31.4] | 23.8 [19.0 to 28.7]
  Week 88: number analyzed (Participants) | 256 | 267
  Week 88 | 29.4 [24.0 to 34.7] | 25.0 [19.9 to 30.0]
  Week 92: number analyzed (Participants) | 247 | 266
  Week 92 | 27.7 [22.2 to 33.1] | 27.3 [22.1 to 32.6]
  Week 96: number analyzed (Participants) | 249 | 258
  Week 96 | 28.0 [22.6 to 33.3] | 26.7 [21.7 to 31.8]
  Week 100: number analyzed (Participants) | 248 | 258
  Week 100 | 27.3 [22.0 to 32.7] | 24.4 [19.5 to 29.3]
  Week 104: number analyzed (Participants) | 250 | 263
  Week 104 | 27.9 [22.5 to 33.3] | 23.9 [18.9 to 28.8]
  Week 108: number analyzed (Participants) | 246 | 256
  Week 108 | 27.3 [21.9 to 32.6] | 24.2 [19.3 to 29.1]
  Week 112: number analyzed (Participants) | 247 | 259
  Week 112 | 26.9 [21.6 to 32.1] | 25.5 [20.4 to 30.6]

17. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/40 or Better (BCVA ≥69 Letters) in the Study Eye Averaged Over Weeks 40, 44, and 48
Description: BCVA was measured on the ETDRS chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity. For each participant, an average BCVA value was calculated across the three visits, and this averaged value was used to determine if the endpoint was met. The results were summarized as the percentage of participants per treatment arm who met the endpoint. The weighted estimates of the percentage of participants were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (<69 letters vs. ≥69 letters), baseline LLD (≥33 letters and <33 letters), and region (U.S. and Canada vs. rest of the world). Treatment policy strategy and hypothetical strategy were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded. 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: Baseline, average of Weeks 40, 44, and 48
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 292 | 300
Percentage of participants | 56.4 [51.5 to 61.4] | 57.0 [51.9 to 62.1]
Statistical Analysis 1: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Treatment Difference in CMH Weighted Percentages at Weeks 40-48; Test type: Other; Difference in CMH Weighted Percentage = -0.5, 95% CI 2-sided [-7.7 to 6.6] — The treatment difference in CMH weighted percentage of participants achieving BCVA ≥69 letters is the calculated difference of Arm A: Faricimab and Arm B: Aflibercept

18. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/40 or Better (BCVA ≥69 Letters) in the Study Eye Over Time
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity. The weighted percentage of participants was based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (<69 letters vs. ≥69 letters), baseline LLD (≥33 letters and <33 letters), and region (U.S. and Canada vs. rest of the world; Asia and rest of the world were combined). Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. Invalid BCVA values were excluded from analysis. 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 334 | 337
Percentage of participants
  Week 4: number analyzed (Participants) | 327 | 331
  Week 4 | 52.8 [48.4 to 57.2] | 50.5 [46.4 to 54.7]
  Week 8: number analyzed (Participants) | 325 | 325
  Week 8 | 54.5 [49.9 to 59.1] | 50.7 [46.3 to 55.1]
  Week 12: number analyzed (Participants) | 322 | 326
  Week 12 | 58.3 [53.7 to 62.9] | 53.4 [48.8 to 58.0]
  Week 16: number analyzed (Participants) | 322 | 320
  Week 16 | 60.4 [55.6 to 65.2] | 53.7 [49.1 to 58.3]
  Week 20: number analyzed (Participants) | 308 | 308
  Week 20 | 59.5 [54.6 to 64.5] | 54.4 [49.6 to 59.1]
  Week 24: number analyzed (Participants) | 278 | 285
  Week 24 | 59.4 [54.3 to 64.5] | 54.4 [49.4 to 59.4]
  Week 28: number analyzed (Participants) | 284 | 276
  Week 28 | 57.5 [52.4 to 62.6] | 59.0 [53.8 to 64.1]
  Week 32: number analyzed (Participants) | 293 | 285
  Week 32 | 57.7 [52.7 to 62.8] | 58.0 [52.8 to 63.1]
  Week 36: number analyzed (Participants) | 286 | 297
  Week 36 | 59.7 [54.8 to 64.7] | 59.6 [54.5 to 64.7]
  Week 40: number analyzed (Participants) | 287 | 291
  Week 40 | 57.5 [52.4 to 62.7] | 58.0 [52.8 to 63.1]
  Week 44: number analyzed (Participants) | 278 | 274
  Week 44 | 59.9 [54.8 to 65.0] | 59.4 [54.1 to 64.7]
  Week 48: number analyzed (Participants) | 273 | 279
  Week 48 | 58.9 [53.7 to 64.1] | 58.1 [52.7 to 63.6]
  Week 52: number analyzed (Participants) | 272 | 278
  Week 52 | 61.0 [55.8 to 66.1] | 57.4 [52.0 to 62.9]
  Week 56: number analyzed (Participants) | 273 | 279
  Week 56 | 59.0 [53.8 to 64.2] | 55.9 [50.5 to 61.3]
  Week 60: number analyzed (Participants) | 268 | 276
  Week 60 | 57.9 [52.4 to 63.4] | 56.8 [51.4 to 62.2]
  Week 64: number analyzed (Participants) | 253 | 276
  Week 64 | 62.5 [57.1 to 67.9] | 57.7 [52.3 to 63.0]
  Week 68: number analyzed (Participants) | 260 | 269
  Week 68 | 61.0 [55.6 to 66.4] | 59.3 [54.0 to 64.6]
  Week 72: number analyzed (Participants) | 262 | 274
  Week 72 | 59.5 [54.0 to 65.0] | 57.3 [52.0 to 62.6]
  Week 76: number analyzed (Participants) | 255 | 260
  Week 76 | 58.4 [52.9 to 63.9] | 55.3 [49.9 to 60.6]
  Week 80: number analyzed (Participants) | 254 | 268
  Week 80 | 56.8 [51.2 to 62.4] | 55.5 [50.1 to 60.9]
  Week 84: number analyzed (Participants) | 257 | 270
  Week 84 | 57.6 [52.1 to 63.1] | 58.0 [52.6 to 63.3]
  Week 88: number analyzed (Participants) | 256 | 267
  Week 88 | 59.1 [53.5 to 64.8] | 54.1 [48.5 to 59.7]
  Week 92: number analyzed (Participants) | 247 | 266
  Week 92 | 58.6 [52.9 to 64.2] | 57.8 [52.3 to 63.2]
  Week 96: number analyzed (Participants) | 249 | 258
  Week 96 | 59.3 [53.7 to 64.9] | 58.3 [52.6 to 64.0]
  Week 100: number analyzed (Participants) | 248 | 258
  Week 100 | 58.1 [52.5 to 63.8] | 57.4 [51.9 to 63.0]
  Week 104: number analyzed (Participants) | 250 | 263
  Week 104 | 59.8 [54.2 to 65.5] | 58.0 [52.4 to 63.6]
  Week 108: number analyzed (Participants) | 246 | 256
  Week 108 | 56.4 [50.7 to 62.1] | 56.4 [50.9 to 62.0]
  Week 112: number analyzed (Participants) | 247 | 259
  Week 112 | 56.3 [50.4 to 62.2] | 54.3 [48.6 to 59.9]

19. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/200 or Worse (BCVA ≤38 Letters) in the Study Eye Averaged Over Weeks 40, 44, and 48
Description: as for outcome 4
Time Frame: Baseline, average of Weeks 40, 44, and 48
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 292 | 300
Percentage of participants | 6.4 [3.7 to 9.1] | 6.9 [4.2 to 9.5]
Statistical Analysis 1: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Treatment Difference in CMH Weighted Percentages at Weeks 40-48; Test type: Other; Difference in CMH Weighted Percentage = -0.5, 95% CI 2-sided [-4.2 to 3.3] — The treatment difference in CMH weighted percentage of participants with BCVA ≤38 letters is the calculated difference of Arm A: Faricimab and Arm B: Aflibercept

20. Secondary Outcome: Percentage of Participants With BCVA Snellen Equivalent of 20/200 or Worse (BCVA ≤38 Letters) in the Study Eye Over Time
Description: as for outcome 6
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 334 | 337
Percentage of participants
  Week 4: number analyzed (Participants) | 327 | 331
  Week 4 | 5.5 [3.2 to 7.9] | 5.5 [3.2 to 7.7]
  Week 8: number analyzed (Participants) | 325 | 325
  Week 8 | 5.8 [3.4 to 8.3] | 5.9 [3.6 to 8.2]
  Week 12: number analyzed (Participants) | 322 | 326
  Week 12 | 4.6 [2.5 to 6.8] | 5.6 [3.3 to 7.9]
  Week 16: number analyzed (Participants) | 322 | 320
  Week 16 | 5.8 [3.5 to 8.2] | 6.3 [3.9 to 8.8]
  Week 20: number analyzed (Participants) | 308 | 308
  Week 20 | 5.9 [3.5 to 8.4] | 6.9 [4.3 to 9.5]
  Week 24: number analyzed (Participants) | 278 | 285
  Week 24 | 4.3 [2.0 to 6.6] | 5.9 [3.4 to 8.5]
  Week 28: number analyzed (Participants) | 284 | 276
  Week 28 | 5.4 [3.0 to 7.9] | 5.2 [2.8 to 7.7]
  Week 32: number analyzed (Participants) | 293 | 285
  Week 32 | 6.1 [3.5 to 8.7] | 6.8 [4.2 to 9.4]
  Week 36: number analyzed (Participants) | 286 | 297
  Week 36 | 6.4 [3.7 to 9.1] | 6.7 [4.1 to 9.3]
  Week 40: number analyzed (Participants) | 287 | 291
  Week 40 | 7.1 [4.3 to 9.9] | 8.1 [5.3 to 11.0]
  Week 44: number analyzed (Participants) | 278 | 274
  Week 44 | 7.0 [4.1 to 9.9] | 6.7 [4.0 to 9.3]
  Week 48: number analyzed (Participants) | 273 | 279
  Week 48 | 7.4 [4.4 to 10.4] | 7.8 [4.9 to 10.7]
  Week 52: number analyzed (Participants) | 272 | 278
  Week 52 | 8.1 [5.0 to 11.1] | 9.4 [6.3 to 12.6]
  Week 56: number analyzed (Participants) | 273 | 279
  Week 56 | 6.3 [3.6 to 9.0] | 7.6 [4.7 to 10.5]
  Week 60: number analyzed (Participants) | 268 | 276
  Week 60 | 6.9 [4.0 to 9.8] | 8.7 [5.6 to 11.7]
  Week 64: number analyzed (Participants) | 253 | 276
  Week 64 | 7.8 [4.6 to 11.0] | 9.1 [6.0 to 12.3]
  Week 68: number analyzed (Participants) | 260 | 269
  Week 68 | 7.6 [4.5 to 10.7] | 9.3 [6.2 to 12.5]
  Week 72: number analyzed (Participants) | 262 | 274
  Week 72 | 8.6 [5.4 to 11.8] | 10.7 [7.5 to 13.9]
  Week 76: number analyzed (Participants) | 255 | 260
  Week 76 | 7.9 [4.7 to 11.1] | 10.8 [7.5 to 14.2]
  Week 80: number analyzed (Participants) | 254 | 268
  Week 80 | 8.8 [5.5 to 12.0] | 10.6 [7.2 to 13.9]
  Week 84: number analyzed (Participants) | 257 | 270
  Week 84 | 7.7 [4.6 to 10.8] | 11.0 [7.8 to 14.2]
  Week 88: number analyzed (Participants) | 256 | 267
  Week 88 | 9.5 [6.1 to 12.9] | 11.7 [8.3 to 15.0]
  Week 92: number analyzed (Participants) | 247 | 266
  Week 92 | 9.0 [5.6 to 12.5] | 12.4 [9.0 to 15.7]
  Week 96: number analyzed (Participants) | 249 | 258
  Week 96 | 8.6 [5.3 to 12.0] | 11.7 [8.2 to 15.1]
  Week 100: number analyzed (Participants) | 248 | 258
  Week 100 | 8.3 [5.0 to 11.5] | 11.9 [8.4 to 15.4]
  Week 104: number analyzed (Participants) | 250 | 263
  Week 104 | 9.4 [6.0 to 12.9] | 11.7 [8.3 to 15.1]
  Week 108: number analyzed (Participants) | 246 | 256
  Week 108 | 7.7 [4.5 to 10.9] | 10.4 [7.1 to 13.7]
  Week 112: number analyzed (Participants) | 247 | 259
  Week 112 | 8.2 [4.9 to 11.5] | 11.8 [8.3 to 15.2]

21. Secondary Outcome: Percentage of Participants in the Faricimab Arm on Once Every 8-Weeks, 12-Weeks, or 16-Weeks Treatment Intervals Among Those Completing Week 48
Description: Percentages are based on the number of participants randomized to the faricimab arm who have not discontinued the study at Week 48. The treatment interval at a given visit is defined as the treatment interval decision followed at that visit. The 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: Week 48
Population: The analysis included all participants randomized to the faricimab arm who completed their Week 48 visit.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab
Number analyzed (Participants) | 315
Percentage of participants
  Once Every 8 Weeks | 20.3 [15.9 to 24.8]
  Once Every 12 Weeks | 34.0 [28.7 to 39.2]
  Once Every 16 Weeks | 45.7 [40.2 to 51.2]

22. Secondary Outcome: Percentage of Participants in the Faricimab Arm on Once Every 8-Weeks, 12-Weeks, or 16-Weeks Treatment Intervals Among Those Completing Week 60
Description: Percentages are based on the number of participants randomized to the faricimab arm who have not discontinued the study at Week 60. The treatment interval at a given visit is defined as the treatment interval decision followed at that visit. The 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: Week 60
Population: The analysis included all participants randomized to the faricimab arm who completed their Week 60 visit.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab
Number analyzed (Participants) | 302
Percentage of participants
  Once Every 8 Weeks | 20.2 [15.7 to 24.7]
  Once Every 12 Weeks | 33.4 [28.1 to 38.8]
  Once Every 16 Weeks | 46.4 [40.7 to 52.0]

23. Secondary Outcome: Percentage of Participants in the Faricimab Arm on Once Every 8-Weeks, 12-Weeks, or 16-Weeks Treatment Intervals Among Those Completing Week 112
Description: Percentages are based on the number of participants randomized to the faricimab arm who have not discontinued the study at Week 112. Treatment interval at a given visit is defined as the treatment interval decision followed at that visit. Treatment interval at Week 112 is calculated using data recorded at Week 108. The 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: Weeks 108 and 112
Population: The analysis included all participants randomized to the faricimab arm who completed their Week 112 visit.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab
Number analyzed (Participants) | 271
Percentage of participants
  Once Every 8 Weeks | 25.8 [20.6 to 31.0]
  Once Every 12 Weeks | 15.1 [10.9 to 19.4]
  Once Every 16 Weeks | 59.0 [53.2 to 64.9]

24. Secondary Outcome: Number of Study Drug Injections Received in the Study Eye Through Week 48
Time Frame: From Baseline through Week 48
Population: Safety Evaluable Population: all participants who received at least one dose of active study drug (faricimab or aflibercept) in the study eye.
Measure: Median (Full Range); unit: Injections
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 333 | 336
Injections | 6.0 [1 to 8] | 8.0 [1 to 8]

25. Secondary Outcome: Number of Study Drug Injections Received in the Study Eye Through Week 60
Time Frame: From Baseline through Week 60
Population: as for outcome 24
Measure: Median (Full Range); unit: Injections
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 333 | 336
Injections | 7.0 [1 to 10] | 9.0 [1 to 9]

26. Secondary Outcome: Number of Study Drug Injections Received in the Study Eye Through Week 108
Time Frame: From Baseline through Week 108
Population: as for outcome 24
Measure: Median (Full Range); unit: Injections
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 333 | 336
Injections | 10.0 [1 to 16] | 15.0 [1 to 15]

27. Secondary Outcome: Change From Baseline in Central Subfield Thickness in the Study Eye Averaged Over Weeks 40, 44, and 48
Description: Central subfield thickness (CST) was defined as the distance between the internal limiting membrane (ILM) and the retinal pigment epithelium (RPE) using optical coherence tomography (OCT), as assessed by the central reading center. For the Mixed Model of Repeated Measures (MMRM) analysis, the model adjusted for treatment group, visit, visit-by-treatment group interaction, baseline CST (continuous), baseline BCVA (≥74 letters, 73-55 letters, and ≤54 letters), baseline LLD (<33 letters and ≥33 letters), and region (U.S. and Canada, Asia, and the rest of the world). An unstructured covariance structure was used. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were implicitly imputed by MMRM. 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: From Baseline through Week 48
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: microns
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 334 | 337
microns | -136.8 [-142.6 to -131.0] | -129.4 [-135.2 to -123.5]
Statistical Analysis 1: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Treatment Difference in Adjusted Means at Weeks 40-48; Test type: Other; Adjusted mean difference = -7.4, 95% CI 2-sided [-15.7 to 0.8], Standard Error of Mean 4.19 — The treatment difference in adjusted means of change from baseline CST is the calculated difference of Arm A: Faricimab and Arm B: Aflibercept. MMRM adjustments are listed in the outcome measure description

28. Secondary Outcome: Change From Baseline in Central Subfield Thickness in the Study Eye Averaged Over Weeks 52, 56, and 60
Description: as for outcome 27
Time Frame: From Baseline through Week 60
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: microns
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 334 | 337
microns | -134.5 [-140.5 to -128.6] | -135.5 [-141.5 to -129.6]
Statistical Analysis 1: Comparison: Arm A: Faricimab vs Arm B: Aflibercept; Treatment Difference in Adjusted Means at Weeks 52-60; Test type: Other; Adjusted mean difference = 1.0, 95% CI 2-sided [-7.4 to 9.4], Standard Error of Mean 4.26 — [estimate comment as in outcome 27, analysis 1]

29. Secondary Outcome: Change From Baseline in Central Subfield Thickness in the Study Eye Over Time
Description: as for outcome 27
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: microns
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 334 | 337
microns
  Week 4 | -131.7 [-137.9 to -125.4] | -116.3 [-122.5 to -110.1]
  Week 8 | -142.6 [-148.1 to -137.2] | -131.8 [-137.2 to -126.3]
  Week 12 | -149.0 [-154.1 to -143.9] | -136.1 [-141.2 to -131.1]
  Week 16 | -148.7 [-155.1 to -142.3] | -110.4 [-116.8 to -104.0]
  Week 20 | -132.9 [-139.2 to -126.6] | -136.1 [-142.4 to -129.8]
  Week 24 | -128.8 [-135.9 to -121.8] | -115.5 [-122.6 to -108.5]
  Week 28 | -129.1 [-135.5 to -122.8] | -132.5 [-139.0 to -126.1]
  Week 32 | -142.7 [-150.2 to -135.2] | -114.5 [-122.0 to -107.0]
  Week 36 | -132.8 [-138.9 to -126.7] | -139.1 [-145.2 to -133.1]
  Week 40 | -140.8 [-148.0 to -133.7] | -123.9 [-131.0 to -116.7]
  Week 44 | -133.9 [-139.9 to -128.0] | -142.4 [-148.3 to -136.4]
  Week 48 | -138.1 [-145.1 to -131.2] | -126.0 [-132.9 to -119.1]
  Week 52 | -139.9 [-146.2 to -133.6] | -139.6 [-145.9 to -133.3]
  Week 56 | -140.4 [-147.4 to -133.3] | -125.9 [-133.0 to -118.9]
  Week 60 | -124.1 [-131.1 to -117.1] | -143.5 [-150.4 to -136.5]
  Week 64 | -145.4 [-152.4 to -138.4] | -127.8 [-134.7 to -120.9]
  Week 68 | -137.5 [-144.0 to -130.9] | -142.8 [-149.4 to -136.3]
  Week 72 | -139.7 [-147.2 to -132.3] | -132.0 [-139.4 to -124.7]
  Week 76 | -135.3 [-142.2 to -128.3] | -142.8 [-149.8 to -135.9]
  Week 80 | -146.7 [-154.3 to -139.0] | -132.1 [-139.7 to -124.5]
  Week 84 | -141.7 [-148.4 to -135.0] | -143.2 [-149.9 to -136.6]
  Week 88 | -143.9 [-150.7 to -137.2] | -139.3 [-146.0 to -132.6]
  Week 92 | -144.8 [-151.1 to -138.4] | -148.5 [-154.7 to -142.2]
  Week 96 | -147.6 [-154.6 to -140.5] | -139.7 [-146.7 to -132.8]
  Week 100 | -145.7 [-152.7 to -138.7] | -147.1 [-153.9 to -140.2]
  Week 104 | -147.7 [-154.6 to -140.8] | -143.4 [-150.2 to -136.6]
  Week 108 | -141.7 [-148.5 to -134.8] | -151.0 [-157.7 to -144.2]
  Week 112 | -150.1 [-157.1 to -143.1] | -144.3 [-151.3 to -137.4]

30. Secondary Outcome: Percentage of Participants With Absence of Intraretinal Fluid in the Study Eye Over Time
Description: Intraretinal fluid was measured using optical coherence tomography (OCT) in the central subfield (center 1 millimetre [mm]). The weighted estimates of the percentage of participants with absence of intraretinal fluid were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥74 letters, 73-55 letters, and ≤54 letters), baseline LLD (≥33 letters and <33 letters), and region (U.S. and Canada vs. rest of the world). Asia and rest of the world regions were combined due to a small number of enrolled participants. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 104, 108, and 112
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 334 | 337
Percentage of participants
  Week 4: number analyzed (Participants) | 324 | 332
  Week 4 | 89.2 [86.0 to 92.4] | 85.2 [81.6 to 88.8]
  Week 8: number analyzed (Participants) | 321 | 325
  Week 8 | 87.5 [84.1 to 90.9] | 84.3 [80.6 to 88.1]
  Week 12: number analyzed (Participants) | 320 | 323
  Week 12 | 89.3 [86.1 to 92.5] | 85.4 [81.8 to 89.0]
  Week 16: number analyzed (Participants) | 318 | 315
  Week 16 | 89.2 [86.0 to 92.5] | 76.3 [71.8 to 80.8]
  Week 20: number analyzed (Participants) | 307 | 306
  Week 20 | 82.4 [78.3 to 86.5] | 83.4 [79.5 to 87.3]
  Week 24: number analyzed (Participants) | 279 | 284
  Week 24 | 80.5 [75.9 to 85.0] | 77.7 [73.0 to 82.4]
  Week 28: number analyzed (Participants) | 285 | 276
  Week 28 | 76.9 [72.3 to 81.4] | 85.3 [81.3 to 89.2]
  Week 32: number analyzed (Participants) | 291 | 285
  Week 32 | 86.8 [83.1 to 90.6] | 79.1 [74.6 to 83.7]
  Week 36: number analyzed (Participants) | 284 | 295
  Week 36 | 79.9 [75.5 to 84.3] | 83.5 [79.4 to 87.6]
  Week 40: number analyzed (Participants) | 276 | 285
  Week 40 | 82.1 [77.7 to 86.5] | 77.2 [72.5 to 81.9]
  Week 44: number analyzed (Participants) | 273 | 264
  Week 44 | 75.5 [70.6 to 80.3] | 84.9 [80.7 to 89.1]
  Week 48: number analyzed (Participants) | 263 | 267
  Week 48 | 82.1 [77.7 to 86.5] | 74.4 [69.4 to 79.5]
  Week 52: number analyzed (Participants) | 273 | 277
  Week 52 | 83.1 [78.8 to 87.4] | 85.0 [80.9 to 89.1]
  Week 56: number analyzed (Participants) | 271 | 276
  Week 56 | 84.9 [80.8 to 89.1] | 80.3 [75.8 to 84.9]
  Week 60: number analyzed (Participants) | 265 | 264
  Week 60 | 72.9 [67.9 to 77.9] | 82.3 [77.9 to 86.7]
  Week 104: number analyzed (Participants) | 249 | 263
  Week 104 | 80.0 [75.2 to 84.8] | 80.7 [76.1 to 85.4]
  Week 108: number analyzed (Participants) | 243 | 253
  Week 108 | 77.8 [72.9 to 82.7] | 84.7 [80.5 to 88.9]
  Week 112: number analyzed (Participants) | 245 | 256
  Week 112 | 82.3 [77.7 to 86.9] | 76.2 [71.0 to 81.3]

31. Secondary Outcome: Percentage of Participants With Absence of Subretinal Fluid in the Study Eye Over Time
Description: Subretinal fluid was measured using optical coherence tomography (OCT) in the central subfield (center 1 mm). The weighted estimates of the percentage of participants with absence of subretinal fluid were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥74 letters, 73-55 letters, and ≤54 letters), baseline LLD (≥33 letters and <33 letters), and region (U.S. and Canada vs. rest of the world). Asia and rest of the world regions were combined due to a small number of enrolled participants. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 104, 108, and 112
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 334 | 337
Percentage of participants
  Week 4: number analyzed (Participants) | 324 | 332
  Week 4 | 67.8 [62.9 to 72.7] | 58.8 [53.7 to 64.0]
  Week 8: number analyzed (Participants) | 321 | 324
  Week 8 | 84.5 [80.6 to 88.4] | 76.4 [71.9 to 81.0]
  Week 12: number analyzed (Participants) | 321 | 324
  Week 12 | 87.2 [83.6 to 90.8] | 78.5 [74.1 to 82.9]
  Week 16: number analyzed (Participants) | 318 | 316
  Week 16 | 89.6 [86.3 to 92.9] | 59.9 [54.6 to 65.2]
  Week 20: number analyzed (Participants) | 307 | 307
  Week 20 | 75.1 [70.3 to 79.9] | 76.3 [71.6 to 81.0]
  Week 24: number analyzed (Participants) | 279 | 284
  Week 24 | 70.8 [65.6 to 75.9] | 63.9 [58.4 to 69.4]
  Week 28: number analyzed (Participants) | 285 | 276
  Week 28 | 71.1 [65.9 to 76.2] | 78.8 [74.0 to 83.5]
  Week 32: number analyzed (Participants) | 292 | 285
  Week 32 | 82.2 [77.9 to 86.5] | 65.1 [59.6 to 70.6]
  Week 36: number analyzed (Participants) | 285 | 295
  Week 36 | 74.1 [69.2 to 79.1] | 79.9 [75.4 to 84.4]
  Week 40: number analyzed (Participants) | 284 | 288
  Week 40 | 78.5 [73.9 to 83.1] | 67.3 [61.9 to 72.7]
  Week 44: number analyzed (Participants) | 277 | 274
  Week 44 | 69.6 [64.3 to 74.9] | 78.0 [73.1 to 82.8]
  Week 48: number analyzed (Participants) | 268 | 279
  Week 48 | 75.7 [70.7 to 80.8] | 65.8 [60.4 to 71.1]
  Week 52: number analyzed (Participants) | 273 | 278
  Week 52 | 80.6 [76.0 to 85.2] | 79.9 [75.3 to 84.5]
  Week 56: number analyzed (Participants) | 271 | 276
  Week 56 | 79.0 [74.3 to 83.7] | 70.1 [64.7 to 75.4]
  Week 60: number analyzed (Participants) | 267 | 274
  Week 60 | 67.7 [62.2 to 73.2] | 77.5 [72.6 to 82.3]
  Week 104: number analyzed (Participants) | 249 | 261
  Week 104 | 79.3 [74.5 to 84.2] | 74.9 [69.7 to 80.1]
  Week 108: number analyzed (Participants) | 245 | 253
  Week 108 | 79.6 [74.6 to 84.6] | 77.4 [72.4 to 82.5]
  Week 112: number analyzed (Participants) | 245 | 256
  Week 112 | 80.9 [76.1 to 85.7] | 73.1 [67.7 to 78.4]

32. Secondary Outcome: Percentage of Participants With Absence of Intraretinal Fluid and Subretinal Fluid in the Study Eye Over Time
Description: Intraretinal fluid and subretinal fluid were measured using optical coherence tomography (OCT) in the central subfield (center 1 millimetre [mm]). The weighted estimates of the percentage of participants with absence of intraretinal and subretinal fluid were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥74 letters, 73-55 letters, and ≤54 letters), baseline LLD (≥33 letters and <33 letters), and region (U.S. and Canada vs. rest of the world). Asia and rest of the world regions were combined due to a small number of enrolled participants. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 104, 108, and 112
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 334 | 337
Percentage of participants
  Week 4: number analyzed (Participants) | 323 | 332
  Week 4 | 60.8 [55.7 to 66.0] | 49.0 [43.8 to 54.2]
  Week 8: number analyzed (Participants) | 321 | 324
  Week 8 | 74.5 [69.9 to 79.2] | 63.1 [58.0 to 68.2]
  Week 12: number analyzed (Participants) | 319 | 323
  Week 12 | 77.4 [72.9 to 81.9] | 66.3 [61.4 to 71.3]
  Week 16: number analyzed (Participants) | 318 | 315
  Week 16 | 78.8 [74.4 to 83.2] | 44.0 [38.6 to 49.4]
  Week 20: number analyzed (Participants) | 307 | 306
  Week 20 | 64.7 [59.4 to 70.0] | 62.2 [56.9 to 67.4]
  Week 24: number analyzed (Participants) | 279 | 284
  Week 24 | 57.2 [51.6 to 62.9] | 48.9 [43.2 to 54.6]
  Week 28: number analyzed (Participants) | 285 | 276
  Week 28 | 54.8 [49.2 to 60.5] | 66.9 [61.5 to 72.3]
  Week 32: number analyzed (Participants) | 292 | 285
  Week 32 | 71.9 [66.8 to 77.0] | 51.2 [45.5 to 56.9]
  Week 36: number analyzed (Participants) | 285 | 295
  Week 36 | 59.4 [53.7 to 65.1] | 66.6 [61.3 to 71.9]
  Week 40: number analyzed (Participants) | 278 | 286
  Week 40 | 64.8 [59.3 to 70.3] | 52.1 [46.3 to 57.9]
  Week 44: number analyzed (Participants) | 275 | 266
  Week 44 | 51.4 [45.6 to 57.2] | 65.5 [59.8 to 71.1]
  Week 48: number analyzed (Participants) | 264 | 268
  Week 48 | 63.3 [57.6 to 68.9] | 47.1 [41.3 to 52.9]
  Week 52: number analyzed (Participants) | 273 | 277
  Week 52 | 68.4 [63.0 to 73.8] | 68.4 [63.1 to 73.8]
  Week 56: number analyzed (Participants) | 271 | 276
  Week 56 | 67.8 [62.3 to 73.3] | 55.3 [49.4 to 61.1]
  Week 60: number analyzed (Participants) | 266 | 267
  Week 60 | 48.6 [42.7 to 54.4] | 62.4 [56.7 to 68.2]
  Week 104: number analyzed (Participants) | 249 | 261
  Week 104 | 63.0 [57.0 to 68.9] | 59.0 [53.1 to 65.0]
  Week 108: number analyzed (Participants) | 243 | 253
  Week 108 | 60.7 [54.7 to 66.8] | 63.6 [57.8 to 69.4]
  Week 112: number analyzed (Participants) | 244 | 256
  Week 112 | 65.9 [60.0 to 71.8] | 54.5 [48.4 to 60.6]

33. Secondary Outcome: Percentage of Participants With Absence of Pigment Epithelial Detachment in the Study Eye Over Time
Description: Pigment epithelial detachment was measured using optical coherence tomography (OCT) in the central subfield (center 1 mm). The weighted estimates of the percentage of participants with absence of pigment epithelial detachment were based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (≥74 letters, 73-55 letters, and ≤54 letters), baseline LLD (≥33 letters and <33 letters), and region (U.S. and Canada vs. rest of the world). Asia and rest of the world regions were combined due to a small number of enrolled participants. Treatment policy strategy (i.e., all observed values used) and hypothetical strategy (i.e., all values censored after the occurrence of the intercurrent event) were applied to non-COVID-19 related and COVID-19 related intercurrent events, respectively. Missing data were not imputed. 95% confidence interval (CI) is a rounding of 95.03% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 104, 108, and 112
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 334 | 337
Percentage of participants
  Week 4: number analyzed (Participants) | 325 | 332
  Week 4 | 5.3 [2.9 to 7.6] | 4.9 [2.6 to 7.2]
  Week 8: number analyzed (Participants) | 320 | 325
  Week 8 | 3.5 [1.5 to 5.5] | 4.3 [2.1 to 6.5]
  Week 12: number analyzed (Participants) | 322 | 325
  Week 12 | 2.9 [1.0 to 4.7] | 2.1 [0.6 to 3.7]
  Week 16: number analyzed (Participants) | 318 | 316
  Week 16 | 1.6 [0.2 to 3.0] | 4.4 [2.2 to 6.6]
  Week 20: number analyzed (Participants) | 306 | 309
  Week 20 | 2.4 [0.7 to 4.1] | 3.9 [1.8 to 6.1]
  Week 24: number analyzed (Participants) | 279 | 285
  Week 24 | 3.3 [1.2 to 5.4] | 4.2 [1.9 to 6.6]
  Week 28: number analyzed (Participants) | 285 | 276
  Week 28 | 2.9 [1.0 to 4.8] | 5.8 [3.1 to 8.5]
  Week 32: number analyzed (Participants) | 292 | 285
  Week 32 | 3.4 [1.4 to 5.5] | 3.6 [1.4 to 5.7]
  Week 36: number analyzed (Participants) | 285 | 295
  Week 36 | 4.3 [1.9 to 6.6] | 6.4 [3.7 to 9.2]
  Week 40: number analyzed (Participants) | 284 | 291
  Week 40 | 7.8 [4.7 to 10.9] | 9.9 [6.5 to 13.3]
  Week 44: number analyzed (Participants) | 277 | 273
  Week 44 | 3.6 [1.5 to 5.8] | 8.8 [5.5 to 12.2]
  Week 48: number analyzed (Participants) | 270 | 279
  Week 48 | 3.4 [1.3 to 5.5] | 7.7 [4.6 to 10.7]
  Week 52: number analyzed (Participants) | 273 | 278
  Week 52 | 2.3 [0.5 to 4.1] | 3.5 [1.4 to 5.7]
  Week 56: number analyzed (Participants) | 271 | 276
  Week 56 | 2.6 [0.7 to 4.5] | 5.8 [3.0 to 8.5]
  Week 60: number analyzed (Participants) | 267 | 274
  Week 60 | 4.2 [1.8 to 6.5] | 6.4 [3.6 to 9.2]
  Week 104: number analyzed (Participants) | 249 | 263
  Week 104 | 3.7 [1.4 to 6.0] | 4.9 [2.3 to 7.6]
  Week 108: number analyzed (Participants) | 243 | 252
  Week 108 | 3.1 [0.9 to 5.4] | 7.5 [4.2 to 10.7]
  Week 112: number analyzed (Participants) | 246 | 256
  Week 112 | 4.0 [1.6 to 6.4] | 8.0 [4.7 to 11.2]

34. Secondary Outcome: Percentage of Participants With Absence of Intraretinal Cysts in the Study Eye Over Time
Time Frame: Up to 112 weeks
Population: The percentage of participants with absence of intraretinal cysts over time was planned but it was not evaluated (i.e., 0 participants analyzed) because the absence of intraretinal fluid and the absence of intraretinal cysts are described by the same variable during reading center grading.
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: Change From Baseline in Total Area of Choroidal Neovascularization Lesion in the Study Eye at Week 48
Description: The total area of the choroidal neovascularization lesion in the study eye was evaluated by a central reading center using fundus fluorescein angiography (FFA). Assessments were censored following COVID-19 related intercurrent events. Baseline was defined as the last available measurement obtained on or prior to randomization.
Time Frame: Baseline and Week 48
Population: ITT Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization. Only participants with non-missing, valid assessments at Baseline and Week 48 were included in this analysis.
Measure: Mean (Standard Deviation); unit: millimetres squared (mm^2)
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 237 | 248
millimetres squared (mm^2) | 0.0 (4.5) | 0.4 (4.8)

36. Secondary Outcome: Change From Baseline in Total Area of Choroidal Neovascularization Lesion in the Study Eye at Week 112
Description: as for outcome 35
Time Frame: Baseline and Week 112
Population: ITT Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization. Only participants with non-missing, valid assessments at Baseline and Week 112 were included in this analysis.
Measure: Mean (Standard Deviation); unit: millimetres squared (mm^2)
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 225 | 236
millimetres squared (mm^2) | 1.2 (4.6) | 1.6 (5.0)

37. Secondary Outcome: Change From Baseline in Total Area of Choroidal Neovascularization Leakage in the Study Eye at Week 48
Description: The total area of choroidal neovascularization leakage in the study eye was evaluated by a central reading center using fundus fluorescein angiography (FFA). Assessments were censored following COVID-19 related intercurrent events. Baseline was defined as the last available measurement obtained on or prior to randomization.
Time Frame: Baseline and Week 48
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: millimetres squared (mm^2)
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 243 | 246
millimetres squared (mm^2) | -3.8 (6.9) | -3.0 (6.9)

38. Secondary Outcome: Change From Baseline in Total Area of Choroidal Neovascularization Leakage in the Study Eye at Week 112
Description: as for outcome 37
Time Frame: Baseline and Week 112
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: millimetres squared (mm^2)
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 222 | 233
millimetres squared (mm^2) | -5.4 (5.7) | -5.0 (6.4)

39. Secondary Outcome: Percentage of Participants With at Least One Adverse Event
Description: This analysis of adverse events (AEs) includes both ocular and non-ocular (systemic) AEs. Multiple occurrences of the same AE in one individual are counted only once. Investigators sought information on AEs at each contact with the participants. All AEs were recorded and the investigator made an assessment of seriousness, severity, and causality of each AE. AEs of special interest included the following: Cases of potential drug-induced liver injury that include an elevated ALT or AST in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's Law; Suspected transmission of an infectious agent by the study drug; Sight-threatening AEs that cause a drop in visual acuity (VA) score ≥30 letters lasting more than 1 hour, require surgical or medical intervention to prevent permanent loss of sight, or are associated with severe intraocular inflammation (IOI).
Time Frame: From first dose of study drug through end of study (up to 112 weeks)
Population: as for outcome 24
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 333 | 336
Percentage of participants
  Adverse Event (AE) | 88.3 | 89.3
  Serious AE (SAE) | 24.0 | 27.7
  AE Leading to Withdrawal from Study Treatment | 3.6 | 2.7
  AE of Special Interest (AESI) | 4.8 | 6.8

40. Secondary Outcome: Percentage of Participants With at Least One Ocular Adverse Event in the Study Eye or the Fellow Eye
Description: This analysis of adverse events (AEs) only includes ocular AEs, which are categorized as having occurred either in the study eye or the fellow eye. Multiple occurrences of the same AE in one individual are counted only once. Investigators sought information on AEs at each contact with the participants. All AEs were recorded and the investigator made an assessment of seriousness, severity, and causality of each AE. Ocular AEs of special interest included the following: Suspected transmission of an infectious agent by the study drug; Sight-threatening AEs that cause a drop in visual acuity (VA) score ≥30 letters lasting more than 1 hour, require surgical or medical intervention to prevent permanent loss of sight, or are associated with severe intraocular inflammation (IOI).
Time Frame: From first dose of study drug through end of study (up to 112 weeks)
Population: as for outcome 24
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 333 | 336
Percentage of participants
  Study Eye: Adverse Event (AE) | 55.0 | 56.5
  Study Eye: Serious AE (SAE) | 4.2 | 3.9
  Study Eye: AE Leading to Withdrawal from Treatment | 1.8 | 0.6
  Study Eye: Treatment-related AE | 4.2 | 2.7
  Study Eye: Treatment-related SAE | 1.2 | 0.0
  Study Eye: AE of Special Interest (AESI) | 3.6 | 3.9
  Study Eye: AESI, Drop in VA Score ≥30 Letters | 2.7 | 3.0
  Study Eye: AESI, Associated with Severe IOI | 0.3 | 0.3
  Study Eye: AESI, Intervention Req. to Prevent Permanent Vision Loss | 0.6 | 0.6
  Fellow Eye: AE | 39.3 | 44.3
  Fellow Eye: SAE | 1.2 | 3.3
  Fellow Eye: AESI | 1.2 | 3.0
  Fellow Eye: AESI, Drop in VA Score ≥30 Letters | 0.9 | 2.1
  Fellow Eye: AESI, Intervention Req. to Prevent Permanent Vision Loss | 0.3 | 0.9

41. Secondary Outcome: Percentage of Participants With at Least One Non-Ocular Adverse Event
Description: This analysis of adverse events (AEs) only includes non-ocular (systemic) AEs. Multiple occurrences of the same AE in one individual are counted only once. Investigators sought information on AEs at each contact with the participants. All AEs were recorded and the investigator made an assessment of seriousness, severity, and causality of each AE. The non-ocular AE of special interest was: Cases of potential drug-induced liver injury that include an elevated ALT or AST in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's Law.
Time Frame: From first dose of study drug through end of study (up to 112 weeks)
Population: as for outcome 24
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
Number analyzed (Participants) | 333 | 336
Percentage of participants
  Adverse Event (AE) | 75.7 | 72.9
  Serious AE (SAE) | 19.8 | 22.6
  AE Leading to Withdrawal from Study Treatment | 1.8 | 2.1
  AE of Special Interest (AESI) | 0.0 | 0.3

42. Secondary Outcome: Plasma Concentration of Faricimab Over Time
Description: Faricimab concentration in plasma was determined using a validated immunoassay method.
Time Frame: Pre-dose at Baseline, Weeks 4, 16, 20, 48, 76, and 112
Population: This analysis only includes Arm A participants who received treatment with faricimab in the pharmacokinetic-evaluable population, which includes safety-evaluable participants with at least one plasma sample, provided sufficient dosing information (dose and dosing time) was available. The number of participants analyzed at a given timepoint includes those with an available plasma sample and dosing information at that timepoint.
Measure: Mean (Standard Deviation); unit: micrograms per millilitre (μg/mL)
Arm/Group | Arm A: Faricimab
Number analyzed (Participants) | 333
micrograms per millilitre (μg/mL)
  Baseline: number analyzed (Participants) | 323
  Baseline | 0.0000 (0.0005)
  Week 4: number analyzed (Participants) | 321
  Week 4 | 0.0288 (0.0194)
  Week 16: number analyzed (Participants) | 304
  Week 16 | 0.0337 (0.0266)
  Week 20: number analyzed (Participants) | 296
  Week 20 | 0.0044 (0.0062)
  Week 48: number analyzed (Participants) | 279
  Week 48 | 0.0139 (0.0175)
  Week 76: number analyzed (Participants) | 258
  Week 76 | 0.0057 (0.0109)
  Week 112: number analyzed (Participants) | 248
  Week 112 | 0.0099 (0.0140)

43. Secondary Outcome: Percentage of Participants Who Tested Positive for Treatment-Emergent Anti-Drug Antibodies Against Faricimab During the Study
Description: Anti-drug antibodies (ADAs) against fariciamb were detected in plasma using a validated bridging enzyme-linked immunosorbent assay (ELISA). The percentage of participants with treatment-emergent ADA-positive samples includes post-baseline evaluable participants with at least one treatment-induced (defined as having an ADA-negative sample or missing sample at baseline and any positive post-baseline sample) or treatment-boosted (defined as having an ADA-positive sample at baseline and any positive post-baseline sample with a titer that is equal to or greater than 4-fold baseline titer) ADA-positive sample during the study treatment period.
Time Frame: Pre-dose at Baseline, Weeks 4, 20, 48, 76, and 112
Population: The immunogenicity-analysis population includes all participants randomized to the faricimab arm with at least one determinant ADA assessment. Only those with at least one post-baseline ADA assessment were included in this analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A: Faricimab
Number analyzed (Participants) | 330
Percentage of participants
  Total Treatment-Emergent ADA-Positive | 11.5
  Treatment-Induced ADA-Positive | 11.2
  Treatment-Boosted ADA-Positive | 0.3

ADVERSE EVENTS:
Time Frame: From first dose of study drug through end of study (up to 112 weeks)
Description: Adverse events (AEs) are reported for the safety population, which includes all participants who received at least one injection of active study drug (faricimab or aflibercept) in the study eye. For ocular AEs, the number of participants and events reported per term are combined totals of AEs that occurred in the study eye or the fellow eye.
Arm/Group | Arm A: Faricimab | Arm B: Aflibercept
All-Cause Mortality (participants affected / at risk) | 13/333 | 7/336
Serious Adverse Events (participants affected / at risk) | 80/333 | 93/336
Other Adverse Events (participants affected / at risk) | 211/333 | 200/336
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Faricimab (N=333) | Arm B: Aflibercept (N=336)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 5 (6) | 4 (4)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 3 (3) | 1 (1)
Mitral valve prolapse (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis constrictive (Cardiac disorders) | 1 (1) | 0 (0)
Age-related macular degeneration (Eye disorders) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 2 (2) | 5 (5)
Neovascular age-related macular degeneration (Eye disorders) | 1 (1) | 9 (11)
Retinal pigment epithelial tear (Eye disorders) | 2 (2) | 0 (0)
Rhegmatogenous retinal detachment (Eye disorders) | 1 (1) | 2 (4)
Subretinal fibrosis (Eye disorders) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (2)
Asthenia (General disorders) | 0 (0) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 2 (2)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1) | 1 (1)
Biliary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 5 (5) | 4 (4)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 5 (5)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Systemic bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Viral uveitis (Infections and infestations) | 1 (1) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hair follicle tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (3) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (2) | 2 (3)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Dry age-related macular degeneration (Eye disorders) | 1 (1) | 0 (0)
Lens dislocation (Eye disorders) | 1 (1) | 0 (0)
Macular degeneration (Eye disorders) | 2 (2) | 0 (0)
Retinal degeneration (Eye disorders) | 0 (0) | 1 (1)
Retinal depigmentation (Eye disorders) | 1 (1) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 1 (1)
Tractional retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Hernia (General disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Cellulitis (Infections and infestations) | 1 (2) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Endophthalmitis (Infections and infestations) | 3 (3) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 1 (1)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intraocular pressure increased (Investigations) | 0 (0) | 2 (2)
Staphylococcus test positive (Investigations) | 0 (0) | 1 (1)
Magnesium deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tracheal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Intensive care unit acquired weakness (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0)
Internal haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Faricimab (N=333) | Arm B: Aflibercept (N=336)
Conjunctival haemorrhage (Eye disorders) | 36 (44) | 33 (40)
Neovascular age-related macular degeneration (Eye disorders) | 65 (85) | 63 (77)
Nasopharyngitis (Infections and infestations) | 23 (27) | 35 (42)
Cataract (Eye disorders) | 27 (41) | 36 (47)
Dry eye (Eye disorders) | 18 (27) | 24 (42)
Eye pain (Eye disorders) | 14 (17) | 18 (25)
Vitreous detachment (Eye disorders) | 19 (23) | 21 (33)
Vitreous floaters (Eye disorders) | 23 (30) | 12 (17)
Urinary tract infection (Infections and infestations) | 26 (37) | 23 (27)
Fall (Injury, poisoning and procedural complications) | 20 (29) | 20 (24)
Intraocular pressure increased (Investigations) | 17 (23) | 14 (22)
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 (25) | 19 (20)
Hypertension (Vascular disorders) | 24 (25) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/87/NCT03823287/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT03823287/SAP_001.pdf